CLINICAL TRIAL: NCT03728881
Title: Non-Inferiority Trial Comparing Immunogenicity From 1-Dose of Bivalent HPV Vaccine in Girls to 3-Doses of Quadrivalent Vaccine in Women: The PRIMAVERA-ESCUDDO Trial ("Puente de Respuesta Inmunológica Para Mejorar el Acceso a Vacunas y Erradicar el Cancer")
Brief Title: Single Dose of Cervarix Vaccine in Girls or Three Doses of Gardasil Vaccine in Women for the Prevention of Human Papillomavirus Infection, the PRIMAVERA-ESCUDDO Trial
Acronym: PRIMAVERA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Cancer Research UK (Other); Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NCI-2020-07432; NCI-2020-07432 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 19-C-N009 (Other: National Cancer Institute)
Record Dates: First submitted 2018-11-01; First posted 2018-11-02 (Actual); Results first posted 2025-07-20 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Human Papillomavirus-Related Cervical Carcinoma
Keywords: HPV vaccine; Single dose HPV vaccination
MeSH Terms: interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18; human papillomavirus vaccine, L1 type 16, 18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Girls (1D Cervarix®) (Experimental): Participants 9-14 years old receive Cervarix IM at baseline.
  Interventions: Biological: Recombinant Human Papillomavirus Bivalent Vaccine
- Women (3D Gardasil-4®) (Active Comparator): Participants 18-25 years old receive Gardasil IM at baseline and at 2 and 6 months in the absence of unacceptable toxicity.
  Interventions: Biological: Quadrivalent Human Papillomavirus (types 6, 11, 16, 18) Recombinant Vaccine

INTERVENTIONS:
Biological: Quadrivalent Human Papillomavirus (types 6, 11, 16, 18) Recombinant Vaccine — Given IM
  Other Names: Gardasil; Quadrivalent HPV [Type 6, 11, 16 and 18] L1 Virus-Like Particle vaccine; quadrivalent human papillomavirus (types 6, 11, 16, and 18) recombinant vaccine; Recombinant Human Papillomavirus (HPV) Quadrivalent Vaccine; V501
  Arms: Women (3D Gardasil-4®)
Biological: Recombinant Human Papillomavirus Bivalent Vaccine — Given IM
  Other Names: Cervarix; GSK-580299; HPV 16/18 L1 VLP/AS04 VAC; HPV-16/18 VLP/AS04 Vaccine; Human Papillomavirus 16/18 L1 Virus-Like Particle/AS04 Vaccine; Human Papillomavirus Bivalent Types 16 and 18 Vaccine, Recombinant; Human Papillomavirus Vaccine L1 16,18; Human Papillomavirus Vaccine, L1 Type 16, 18; Recombinant HPV Bivalent Vaccine
  Arms: Girls (1D Cervarix®)

SUMMARY:
This phase IIIb trial compares a single dose of the Cervarix vaccine in girls to 3 doses of the Gardasil vaccine in young women for the prevention of human papillomavirus (HPV) infection. Cervarix is a vaccine used to prevent cervical cancer caused by HPV types 16 and 18. Gardasil is vaccine used to prevent cervical, vulvar, and vaginal cancer caused by HPV types 16 and 18 and genital warts caused by HPV types 6 and 11. Giving only one dose of the Cervarix vaccine in girls may work the same as 3 doses of the Gardasil vaccine in young women in preventing HPV infection and ultimately, cervical and other HPV-related cancers. Currently, many women around the world cannot get HPV vaccines because they are too expensive. If this trial can show one dose given to young girls is enough to prevent cancer, more girls might be able to get the vaccine.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To demonstrate that the immunogenicity (as determined by enzyme-linked immunosorbent assay [ELISA]) of a single dose of recombinant human papillomavirus bivalent vaccine (Cervarix) in 9-14 year old girls is non-inferior to the immunogenicity of three doses of quadrivalent human papillomavirus (types 6, 11, 16, 18) recombinant vaccine (Gardasil), administered at 0, 2, and 6 months, in 18-25 year old women 36 months after initial vaccination, with an interim analysis at 24 months after initial vaccination.

SECONDARY OBJECTIVES:

I. To compare the distribution of HPV -16 and HPV-18 antibodies levels, assessed at 24 and 36 months after initial vaccination, following a single dose of Cervarix in 9-14 year old girls and three doses of Gardasil, administered at 0, 2, and 6 months, in 18-25 year old women.

II. To compare rates of seroconversion based on HPV-16 and HPV-18 antibody levels, assessed at 24 and 36 months after initial vaccination, following a single dose of Cervarix in 9-14 year old girls and three doses of Gardasil, administered at 0, 2, and 6 months, in 18-25 year old women.

III. To compare geometric mean titers (GMTs), distributions, and seroconversion rates for HPV-16 and HPV-18 antibodies, assessed at 24 and 36 months after initial vaccination, following a single dose of Cervarix in 9-11 year old girls and three doses of Gardasil, administered at 0, 2, and 6 months, in 18-25 year old women; to perform a similar comparison restricting to 12-14 year old girls.

IV. To compare GMTs, distributions, and seroconversion rates for HPV-16 and HPV-18 antibodies, assessed at 1-month after vaccination and 1-year after vaccination, following a single dose of Cervarix in 9-10 year old girls and a single dose of Cervarix in 11-14 year old girls.

V. To evaluate whether baseline variables (e.g. geographic district, initial antibody levels, date of vaccination) are associated with GMTs, distributions, and seroconversion rates for HPV16 and HPV-18 antibodies, assessed at 24 and 36 months after initial vaccination.

OUTLINE: Participants are assigned to 1 of 2 groups.

GROUP I: Participants 9-14 years old receive Cervarix intramuscularly (IM) at baseline.

GROUP II: Participants 18-25 years old receive Gardasil IM at baseline and at 2 and 6 months in the absence of unacceptable toxicity.

After completion of trial vaccine dose(s), participants are followed up at 1, 12, 24, and 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Aged between:

  * 9 and 14 years inclusive for Cervarix group
  * 18 and 25 years inclusive for Gardasil group
* Living in the study area without plans to move outside the country in the next six months
* Able to communicate with study personnel
* Able and willing to provide a blood sample
* Willing to permit export of blood samples to the United States
* Willing to participate in the study and:

  * If Cervarix group and less than 12 years old, receive study information and be supported in study participation by at least one of parent (or guardian), who is willing to sign the informed consent document
  * If Cervarix group and 12 years old or older, sign the informed assent and be supported in study participation by at least one parent (or guardian), who is willing to sign the informed consent document
  * If Gardasil group, sign the informed consent
* In good health as determined by a medical history (physical exam will be conducted if necessary per the doctor's criterion)

Exclusion Criteria:

* They have a diagnosis of an autoimmune, degenerative, or neurological disease without treatment or adequate control; a progressive or severe neurological disease; a genetic immunodeficiency; or any other serious chronic disease without treatment and / or adequate control that, according to the principal investigator or designee, for which vaccination is contraindicated (NOTE: Potential participants with these conditions can be included after consultation with the external medical advisor of the study or with an appropriate specialist)
* They are allergic to one of the vaccine components, including yeast (if Gardasil group)
* They have received immunoglobulins within 90 days preceding enrollment/vaccination visit
* They are unwilling to provide a blood sample
* Unwilling to permit export of blood samples to the United States
* They have a positive urine pregnancy test result
* They are pregnant
* They are planning to become pregnant
* The clinician determining eligibility in agreement with the principal investigator considers that there is a reason that precludes participation
* They have been vaccinated against HPV
* The participant or her parent/legal guardian, as applicable, does not have an identification document

Ages: 9 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1240 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2024-04-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aimee R Kreimer, Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Agencia Costarricense de Investigaciones Biomédicas (ACIB), Liberia, Guanacaste Province, Costa Rica

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make IPD and related data dictionaries available.

REFERENCES:
- [Background] Cortes B, Ocampo R, Porras C, Liu D, Gail MH, Sierra MS, Herrero R, Lowy DR, Carvajal LJ, Kemp TJ, Fantin R, Schussler J, Hildesheim A, Sampson JN, Pinto LA, Schiller JT, Kreimer AR. Human papillomavirus (HPV) type 16 and type 18 antibody concentrations after a single dose of bivalent HPV vaccine in girls aged 9-14 years compared with three doses of quadrivalent HPV vaccine in women aged 18-25 years in Costa Rica (PRIMAVERA): a non-randomised, open-label, immunobridging, non-inferiority trial. Lancet Infect Dis. 2025 Dec;25(12):1314-1324. doi: 10.1016/S1473-3099(25)00284-1. Epub 2025 Jul 16. PMID 40683285

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Multiple methods were used to reach potential participants within the PRIMAVERA catchment area, including publicizing through attending community events, distributing outreach materials in commercial and residential areas, making announcements, and going door-to-door. As needed for potential participants registered away from their residence, in-person verification of potential participants' addresses was conducted to ensure they resided in the catchment area.
Pre-assignment Details: Of 1655 registered individuals (773 girls 9-14 years old and 882 women 18-25 years old), 113 were ineligible (44 girls and 69 women), 184 refused (91 girls and 93 women), and 118 were excluded due to termination of the field effort (18 girls and 100 women). Individuals were ineligible if they could not provide blood, fell outside the eligible age range, resided outside the catchment area, had previously received an HPV vaccination, or had a medical condition that warranted exclusion.
Period: Enrolled and Received 1st Vaccination
Arm/Group | Girls (1D Cervarix®) | Women (3D Gardasil-4®)
Started | 620 | 620
Received All Vaccines Within the ATP Windows (Gardasil® Arm Only) | 0 | 559
No External HPV Vaccination Based on Self-report (Cervarix® Arm Only) | 595 | 0
No External HPV Vaccination Based on HPV6/11 ELISA Results When Available (Cervarix® Arm Only) | 585 | 0
Provided 36-month Blood in ATP Window | 575 | 545
Completed | 575 | 545
Not Completed | 45 | 75
Not completed — Adverse Event | 0 | 1
Not completed — Death | 1 | 1
Not completed — Withdrawal by Subject | 5 | 8
Not completed — Out of Country | 1 | 3
Not completed — No Show | 0 | 1
Not completed — Unable to appoint | 3 | 12
Not completed — Not fully vaccinated during ATP windows | 0 | 49
Not completed — Received HPV vaccination outside study (self-report) | 25 | 0
Not completed — HPV6/11 positive | 10 | 0
Period: ATP Cohort for HPV16 at 36 Months
Arm/Group | Girls (1D Cervarix®) | Women (3D Gardasil-4®)
Started | 575 | 545
Completed | 539 | 366
Not Completed | 36 | 179
Not completed — HPV16 seropositive at baseline | 36 | 179
Period: ATP Cohort for HPV18 at 36 Months
Arm/Group | Girls (1D Cervarix®) | Women (3D Gardasil-4®)
Started | 575 | 545
Completed | 523 | 373
Not Completed | 52 | 172
Not completed — HPV18 seropositive at baseline | 52 | 172

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Girls (1D Cervarix®) | Women (3D Gardasil-4®) | Total
Number analyzed (Participants) | 620 | 620 | 1240
Age, Customized [Count of Participants; unit: Participants]
  Age: 9 years | 72 | 0 | 72
  Age: 10 years | 44 | 0 | 44
  Age: 11 years | 137 | 0 | 137
  Age: 12 years | 126 | 0 | 126
  Age: 13 years | 126 | 0 | 126
  Age: 14 years | 115 | 0 | 115
  Age: 18 years | 0 | 75 | 75
  Age: 19 years | 0 | 98 | 98
  Age: 20 years | 0 | 82 | 82
  Age: 21 years | 0 | 78 | 78
  Age: 22 years | 0 | 82 | 82
  Age: 23 years | 0 | 63 | 63
  Age: 24 years | 0 | 78 | 78
  Age: 25 years | 0 | 64 | 64
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 620 | 620 | 1240
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number Seropositive for HPV16 at 36 Months
Description: Will measure HPV16 specific serum antibody using the HPV type-specific ELISA on serum. For computing proportions seropositive and proportions seroconverting, HPV16 is seropositive if the ELISA concentration is greater than 1.41 IU/mL. Participants whose analysis of the 36-month sample does not generate a valid HPV16 result will be excluded only from the 36-month HPV16 analysis.
Time Frame: 36 months following initial HPV vaccination
Population: The primary cohort for the final analysis of HPV16 includes participants who received the appropriate number of vaccine doses within the specified windows, were initially seronegative for HPV16, underwent blood collection at the 36-month mark, and reported no additional HPV vaccinations outside the study before the 36-month blood collection, as confirmed by self-report or serologic testing for HPV6/HPV11.
Measure: Count of Participants; unit: Participants
Arm/Group | Girls (1D Cervarix®) | Women (3D Gardasil-4®)
Number analyzed (Participants) | 539 | 366
Participants | 538 | 366

2. Primary Outcome: Immunogenicity for HPV16 of One Dose of Bivalent HPV Vaccine (Cervarix) in 9-14 Year Old Girls Compared to Three Doses of Quadrivalent HPV Vaccine (Gardasil), Administered at 0,2 and 6 Months, in 18-25 Year Old Women, 36 Months After Initial Vaccination
Description: Will measure HPV-16 specific serum antibody using the HPV type-specific ELISA on serum. Will estimate the two-sided 99% confidence interval of the GMT ratios for HPV-16 and HPV-18 at 24 months and the two-sided 96% confidence intervals of the GMT ratios for HPV-16 and HPV-18 at 36 months.
Time Frame: 36 months following initial vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: International units (IU/mL)
Arm/Group | Girls (1D Cervarix®) | Women (3D Gardasil-4®)
Number analyzed (Participants) | 538 | 366
International units (IU/mL) | 21.4 [19.7 to 23.3] | 42.9 [38.9 to 47.3]
Statistical Analysis 1: Comparison: Girls (1D Cervarix®) vs Women (3D Gardasil-4®); This procedure controls the overall type one error at 0.05. We are conducting 4 one-sided tests and will spend alpha as follows: 0.005 of the alpha each for HPV16 and for HPV18 at 24 months and 0.02 of the alpha each for HPV16 and for HPV18 at 36 months. The experiment-wise significance level accounting for multiple comparisons is ≤ 0.05 because the null chance of rejection for either HPV16 or HPV18 is ≤0.01 at 24 months by the Bonferroni inequality and ≤0.04 at 36 months; Test type: Non-Inferiority — Let R=GMC1/GMC3 be the ratio of geometric mean concentrations of 1 dose to 3 doses. We reject the noninferiority hypothesis if at 36 months the lower limit of the two-sided 96% confidence interval on R ≥ 0.67 for HPV16. The overall Type 1 error rate for rejecting the null hypotheses for both HPV16 and HPV18 (i.e., declaring noninferiority of the 1D2V) at either time point was controlled at 0.025; GMC Ratio = 0.5, 96% CI 2-sided [0.44 to 0.57] — Generalized estimating equations were used to estimate R and construct confidence intervals

3. Primary Outcome: Number Seropositive for HPV18 at 36 Months
Description: Will measure HPV18 specific serum antibody using the HPV type-specific ELISA on serum. For computing proportions seropositive and proportions seroconverting, HPV18 is seropositive if the ELISA concentration is greater than 1.05 IU/mL. Participants whose analysis of the 36-month sample does not generate a valid HPV18 result will be excluded only from the 36-month HPV18 analysis.
Time Frame: 36 months following initial vaccination
Population: The primary cohort for the final analysis of HPV18 includes participants who received the appropriate number of vaccine doses within the specified windows, were initially seronegative for HPV18, underwent blood collection at the 36-month mark, and reported no additional HPV vaccinations outside the study before the 36-month blood collection, as confirmed by self-report or serologic testing for HPV6/HPV11.
Measure: Count of Participants; unit: Participants
Arm/Group | Girls (1D Cervarix®) | Women (3D Gardasil-4®)
Number analyzed (Participants) | 523 | 373
Participants | 517 | 358

4. Primary Outcome: Immunogenicity for HPV18 of One Dose of Bivalent HPV Vaccine (Cervarix) in 9-14 Year Old Girls Compared to Three Doses of Quadrivalent HPV Vaccine (Gardasil), Administered at 0,2, and 6 Months, in 18-25 Year Old Women, 36 Months After Initial Vaccination
Description: Will measure HPV-18 specific serum antibody using the HPV type-specific ELISA on serum. Will estimate the two-sided 99% confidence interval of the GMT ratios for HPV-16 and HPV-18 at 24 months and the two-sided 96% confidence intervals of the GMT ratios for HPV-16 and HPV-18 at 36 months.
Time Frame: 36 months following initial vaccination
Population: Will measure HPV-18 specific serum antibody using the HPV type-specific ELISA on serum. Will estimate the two-sided 96% confidence intervals of the Geometric Mean Concentration (GMC) ratio for HPV-18 at 36 months.
Measure: Geometric Mean (95% Confidence Interval); unit: International units (IU/mL)
Arm/Group | Girls (1D Cervarix®) | Women (3D Gardasil-4®)
Number analyzed (Participants) | 517 | 358
International units (IU/mL) | 8.0 [7.4 to 8.8] | 7.2 [6.4 to 8.1]
Statistical Analysis 1: Comparison: Girls (1D Cervarix®) vs Women (3D Gardasil-4®); [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority — Let R=GMC1/GMC3 be the ratio of geometric mean concentrations of 1 dose to 3 doses. We reject the noninferiority hypothesis if at 36 months the lower limit of the two-sided 96% confidence interval on R ≥ 0.67 for HPV18. The overall Type 1 error rate for rejecting the null hypotheses for both HPV16 and HPV18 (i.e., declaring noninferiority of the 1D2V) at either time point was controlled at 0.025; Ratio of the GMCs = 1.11, 96% CI 2-sided [0.95 to 1.29] — Generalized estimating equations were used to estimate R and construct confidence intervals

5. Primary Outcome: Number Seropositive for HPV16 at 24 Months
Description: Will measure HPV16 specific serum antibody using the HPV type-specific ELISA on serum. For computing proportions seropositive and proportions seroconverting, HPV16 is seropositive if the ELISA titer is greater than 1.41 IU/mL. Participants whose analysis of the 24-month sample does not generate a valid HPV16 result will be excluded only from the 24-month HPV16 analysis.
Time Frame: 24 months following initial HPV vaccination
Population: The primary cohort for the interim analysis of HPV16 includes participants who received the appropriate number of vaccine doses within the specified windows, were initially seronegative for HPV16, underwent blood collection at the 24-month mark, and reported no additional HPV vaccinations outside the study before the 24-month blood collection, as confirmed by self-report or serologic testing for HPV6/HPV11.
Measure: Count of Participants; unit: Participants
Arm/Group | Girls (1D Cervarix®) | Women (3D Gardasil-4®)
Number analyzed (Participants) | 547 | 371
Participants | 546 | 371

6. Primary Outcome: Immunogenicity for HPV16 of One Dose of Bivalent HPV Vaccine (Cervarix) in 9-14 Year Old Girls Compared to Three Doses of Quadrivalent HPV Vaccine (Gardasil), Administered at 0,2, and 6 Months, in 18-25 Year Old Women, 24 Months After Initial Vaccination
Description: Will measure HPV-16 specific serum antibody using the HPV type-specific enzyme-linked immunoassay (ELISA) on serum. Will estimate the two-sided 99% confidence interval of the geometric mean concentration (GMC) ratio for HPV-16 at 24 months
Time Frame: 24 months following initial vaccination
Population: The primary cohort for the final analysis of HPV16 includes participants who received the appropriate number of vaccine doses within the specified windows, were initially seronegative for HPV16, underwent blood collection at the 36-month mark, and reported no additional HPV vaccinations outside the study before the 24-month blood collection, as confirmed by self-report or serologic testing for HPV6/HPV11.
Measure: Geometric Mean (95% Confidence Interval); unit: International units (IU/mL)
Arm/Group | Girls (1D Cervarix®) | Women (3D Gardasil-4®)
Number analyzed (Participants) | 546 | 371
International units (IU/mL) | 20.6 [19.0 to 22.4] | 48.8 [44.4 to 53.7]
Statistical Analysis 1: Comparison: Girls (1D Cervarix®) vs Women (3D Gardasil-4®); This procedure controls the overall type one error at 0.05. We are conducting 4 one-sided tests and will spend alpha as follows: 0.005 of the alpha each for HPV16 and for HPV18 at 24 months and 0.02 of the alpha each for HPV16 and for HPV18 at 36 months. The experiment-wise significance level accounting for multiple comparisons is ≤0.05 because the null chance of rejection for either HPV16 or HPV18 is ≤0.01 at 24 months by the Bonferroni inequality and ≤0.04 at 36 months; Test type: Non-Inferiority — Let R=GMC1/GMC3 be the ratio of geometric mean concentrations of 1 dose to 3 doses. We reject the noninferiority hypothesis if at 24 months the lower limit of the two-sided 99% confidence interval on R ≥ 0.67 for HPV16. The overall Type 1 error rate for rejecting the null hypotheses for both HPV16 and HPV18 (i.e., declaring noninferiority of the 1D2V) at either time point was controlled at 0.025; GMC Ratio = 0.42, 99% CI 2-sided [0.36 to 0.50] — Generalized estimating equations were used to estimate R and construct confidence intervals

7. Primary Outcome: Number Seropositive for HPV18 at 24 Months
Description: Will measure HPV18 specific serum antibody using the HPV type-specific ELISA on serum. For computing proportions seropositive and proportions seroconverting, HPV18 is seropositive if the ELISA titer is greater than 1.05 IU/mL. Participants whose analysis of the 24-month sample does not generate a valid HPV18 result will be excluded only from the 24-month HPV18 analysis.
Time Frame: 24 months following initial vaccination
Population: The primary cohort for the interim analysis of HPV18 includes participants who received the appropriate number of vaccine doses within the specified windows, were initially seronegative for HPV18, underwent blood collection at the 24-month mark, and reported no additional HPV vaccinations outside the study before the 24-month blood collection, as confirmed by self-report or serologic testing for HPV6/HPV11.
Measure: Count of Participants; unit: Participants
Arm/Group | Girls (1D Cervarix®) | Women (3D Gardasil-4®)
Number analyzed (Participants) | 530 | 376
Participants | 521 | 367

8. Primary Outcome: Immunogenicity for HPV18 of One Dose of Bivalent HPV Vaccine (Cervarix) in 9-14 Year Old Girls Compared to Three Doses of Quadrivalent HPV Vaccine (Gardasil), Administered at 0,2, and 6 Months, in 18-25 Year Old Women, 24 Months After Initial Vaccination
Description: Will measure HPV-18 specific serum antibody using the HPV type-specific ELISA on serum. Will estimate the two-sided 99% confidence interval of the Geometric Mean Concentration (GMC) ratio for HPV-18 at 24 months.
Time Frame: 24 months following initial vaccination
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: International units (IU/mL)
Arm/Group | Girls (1D Cervarix®) | Women (3D Gardasil-4®)
Number analyzed (Participants) | 521 | 367
International units (IU/mL) | 7.9 [0.7 to 8.6] | 8.8 [7.9 to 9.9]
Statistical Analysis 1: Comparison: Girls (1D Cervarix®) vs Women (3D Gardasil-4®); This procedure controls the overall type one error at 0.05. We are conducting 4 one sided tests and will spend alpha as follows: 0.005 of the alpha each for HPV16 and for HPV18 at 24 months and 0.02 of the alpha each for HPV16 and for HPV18 at 36 months. The experiment-wise significance level accounting for multiple comparisons is ≤0.05 because the null chance of rejection for either HPV16 or HPV18 is ≤0.01 at 24 months by the Bonferroni inequality and ≤0.04 at 36 months; Test type: Non-Inferiority — Let R=GMC1/GMC3 be the ratio of geometric mean concentrations of 1 dose to 3 doses. We reject the noninferiority hypothesis if at 24 months the lower limit of the two-sided 99% confidence interval on R ≥ 0.67 for HPV18. The overall Type 1 error rate for rejecting the null hypotheses for both HPV16 and HPV18 (i.e., declaring noninferiority of the 1D2V) at either time point was controlled at 0.025; GMC Ratio = 0.90, 99% CI 2-sided [0.75 to 1.08] — Generalized estimating equations were used to estimate R and construct confidence intervals

9. Secondary Outcome: Comparison of Proportions With Seroconversion Based on HPV16 Antibody Levels Assessed at 36 Months
Description: To compare proportions with seroconversion based on HPV16 antibody levels, assessed at 36 months after initial vaccination, following a single dose of Cervarix in 9-14 year old girls and following three doses of Gardasil, administered at 0, 2, and 6 months, in 18-25 year old women.
Time Frame: 36 months
Measure: Count of Participants; unit: Participants
Arm/Group | Girls (1D Cervarix®) | Women (3D Gardasil-4®)
Number analyzed (Participants) | 539 | 366
Participants | 538 | 366
Statistical Analysis 1: Comparison: Girls (1D Cervarix®) vs Women (3D Gardasil-4®); Test type: Equivalence — We will use a Fisher Exact test to test for the difference of the seroconversion rate between one-dose and three-dose recipients. A p-value under 0.05 will be regarded as significant; p = 1.0, Fisher Exact

10. Secondary Outcome: Comparison of Proportions With Seroconversion Based on HPV18 Antibody Levels Assessed at 36 Months
Description: To compare proportions with seroconversion based on HPV18 antibody levels, assessed at 36 months after initial vaccination, following a single dose of Cervarix in 9-14 year old girls and following three doses of Gardasil, administered at 0, 2, and 6 months, in 18-25 year old women.
Time Frame: 36 month
Measure: Count of Participants; unit: Participants
Arm/Group | Girls (1D Cervarix®) | Women (3D Gardasil-4®)
Number analyzed (Participants) | 523 | 373
Participants | 517 | 358
Statistical Analysis 1: Comparison: Girls (1D Cervarix®) vs Women (3D Gardasil-4®); Test type: Equivalence — [test comment as in outcome 9, analysis 1]; p = 0.006, Fisher Exact

11. Secondary Outcome: Comparison of Proportions With Seroconversion Based HPV16 Antibody Levels at 24 Months
Description: To compare proportions with seroconversion based on HPV16 antibody levels, assessed at 24 months after initial vaccination, following a single dose of Cervarix in 9-14 year old girls and following three doses of Gardasil, administered at 0, 2, and 6 months, in 18-25 year old women.
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Girls (1D Cervarix®) | Women (3D Gardasil-4®)
Number analyzed (Participants) | 547 | 371
Participants | 547 | 371
Statistical Analysis 1: Comparison: Girls (1D Cervarix®) vs Women (3D Gardasil-4®); Test type: Equivalence — [test comment as in outcome 9, analysis 1]; p = 1.0, Fisher Exact

12. Secondary Outcome: Comparison of Proportions With Seroconversion Based on HPV18 Antibody Levels Assessed at 24 Months
Description: To compare proportions with seroconversion based on HPV18 antibody levels, assessed at 24 months after initial vaccination, following a single dose of Cervarix in 9-14 year old girls and following three doses of Gardasil, administered at 0, 2, and 6 months, in 18-25 year old women.
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Girls (1D Cervarix®) | Women (3D Gardasil-4®)
Number analyzed (Participants) | 530 | 376
Participants | 521 | 367
Statistical Analysis 1: Comparison: Girls (1D Cervarix®) vs Women (3D Gardasil-4®); Test type: Equivalence — [test comment as in outcome 9, analysis 1]; p = 0.48, Fisher Exact

13. Secondary Outcome: Comparison of Distribution of HPV16 Antibodies Levels Assessed at 36 Months
Description: Distribution of HPV16 antibodies levels assessed at 36 months following a single dose of Cervarix in 9-14 year old girls compared to distribution of HPV16 antibodies levels assessed at 36 months following three doses of Gardasil, administered at 0, 2, and 6 months, in 18-25 year old women. Shown as medians and ranges by deciles.
Time Frame: 36 months following initial vaccination
Population: as for outcome 1
Measure: Median (Full Range); unit: International units (IU/mL)
Arm/Group | Girls (1D Cervarix®) | Women (3D Gardasil-4®)
Number analyzed (Participants) | 539 | 366
International units (IU/mL)
  Decile 1: number analyzed (Participants) | 54 | 37
  Decile 1 | 4.39 [0.700 to 5.852] | 9.834 [0.700 to 13.625]
  Decile 2: number analyzed (Participants) | 54 | 37
  Decile 2 | 7.613 [5.853 to 9.357] | 17.245 [13.626 to 20.329]
  Decile 3: number analyzed (Participants) | 54 | 36
  Decile 3 | 11.148 [9.358 to 12.952] | 23.906 [20.330 to 27.172]
  Decile 4: number analyzed (Participants) | 54 | 37
  Decile 4 | 14.896 [12.953 to 16.892] | 31.218 [27.173 to 34.459]
  Decile 5: number analyzed (Participants) | 54 | 36
  Decile 5 | 19.790 [16.893 to 21.527] | 39.034 [34.460 to 43.235]
  Decile 6: number analyzed (Participants) | 54 | 37
  Decile 6 | 23.899 [21.528 to 26.399] | 49.061 [43.236 to 53.882]
  Decile 7: number analyzed (Participants) | 54 | 37
  Decile 7 | 32.194 [26.400 to 37.100] | 59.399 [53.883 to 69.789]
  Decile 8: number analyzed (Participants) | 54 | 36
  Decile 8 | 41.001 [37.101 to 45.715] | 78.081 [69.790 to 88.011]
  Decile 9: number analyzed (Participants) | 54 | 37
  Decile 9 | 56.984 [45.716 to 75.071] | 107.219 [88.012 to 140.529]
  Decile 10: number analyzed (Participants) | 53 | 36
  Decile 10 | 119.929 [75.072 to 529.494] | 200.652 [140.260 to 555.910]

14. Secondary Outcome: Comparison of Distribution of HPV18 Antibodies Levels Assessed at 36 Months
Description: Distribution of HPV18 antibodies levels assessed at 36 months following a single dose of Cervarix in 9-14 year old girls compared to distribution of HPV18 antibodies levels assessed at 36 months following three doses of Gardasil, administered at 0, 2, and 6 months, in 18-25 year old women. Shown in medians and ranges by deciles.
Time Frame: 36 months
Population: as for outcome 3
Measure: Median (Full Range); unit: International units (IU/mL)
Arm/Group | Girls (1D Cervarix®) | Women (3D Gardasil-4®)
Number analyzed (Participants) | 523 | 373
International units (IU/mL)
  Decile 1: number analyzed (Participants) | 53 | 38
  Decile 1 | 1.511 [0.520 to 2.267] | 1.272 [0.520 to 1.824]
  Decile 2: number analyzed (Participants) | 52 | 37
  Decile 2 | 2.748 [2.268 to 3.498] | 2.163 [1.825 to 2.723]
  Decile 3: number analyzed (Participants) | 52 | 37
  Decile 3 | 4.067 [3.499 to 4.962] | 3.518 [2.724 to 3.885]
  Decile 4: number analyzed (Participants) | 53 | 38
  Decile 4 | 5.509 [4.963 to 6.188] | 4.616 [3.886 to 5.279]
  Decile 5: number analyzed (Participants) | 52 | 37
  Decile 5 | 7.056 [6.189 to 8.040] | 6.156 [5.280 to 7.043]
  Decile 6: number analyzed (Participants) | 52 | 37
  Decile 6 | 9.396 [8.041 to 10.551] | 8.152 [7.004 to 9.681]
  Decile 7: number analyzed (Participants) | 53 | 38
  Decile 7 | 12.468 [10.552 to 14.101] | 11.070 [9.682 to 13.141]
  Decile 8: number analyzed (Participants) | 52 | 37
  Decile 8 | 15.708 [14.102 to 17.605] | 15.030 [13.142 to 17.911]
  Decile 9: number analyzed (Participants) | 52 | 37
  Decile 9 | 22.706 [17.606 to 29.016] | 22.107 [17.912 to 36.612]
  Decile 10: number analyzed (Participants) | 52 | 37
  Decile 10 | 40.538 [29.017 to 369.780] | 49.490 [32.613 to 168.932]

15. Secondary Outcome: Comparison of Distribution of HPV16 Antibodies Levels Assessed at 24 Months
Description: Distribution of HPV16 antibodies levels assessed at 24 months following a single dose of Cervarix in 9-14 year old girls compared to distribution of HPV16 antibodies levels assessed at 24 months following three doses of Gardasil, administered at 0, 2, and 6 months, in 18-25 year old women. Shown as medians and ranges by deciles.
Time Frame: 24 months
Population: as for outcome 5
Measure: Median (Full Range); unit: International units (IU/mL)
Arm/Group | Girls (1D Cervarix®) | Women (3D Gardasil-4®)
Number analyzed (Participants) | 547 | 371
International units (IU/mL)
  Decile 1: number analyzed (Participants) | 55 | 38
  Decile 1 | 4.170 [0.700 to 5.780] | 11.071 [0.700 to 14.744]
  Decile 2: number analyzed (Participants) | 55 | 37
  Decile 2 | 7.226 [5.781 to 9.277] | 19.538 [14.745 to 23.657]
  Decile 3: number analyzed (Participants) | 55 | 37
  Decile 3 | 10.966 [9.278 to 12.390] | 27.914 [23.658 to 30.979]
  Decile 4: number analyzed (Participants) | 54 | 37
  Decile 4 | 14.307 [12.391 to 16.160] | 34.679 [30.980 to 38.266]
  Decile 5: number analyzed (Participants) | 55 | 37
  Decile 5 | 18.022 [16.161 to 20.408] | 41.836 [38.267 to 47.324]
  Decile 6: number analyzed (Participants) | 55 | 37
  Decile 6 | 23.439 [20.409 to 26.986] | 55.290 [47.325 to 63.380]
  Decile 7: number analyzed (Participants) | 54 | 37
  Decile 7 | 30.843 [26.987 to 33.419] | 71.274 [63.381 to 81.015]
  Decile 8: number analyzed (Participants) | 55 | 37
  Decile 8 | 39.221 [33.420 to 46.278] | 92.907 [81.016 to 102.904]
  Decile 9: number analyzed (Participants) | 55 | 37
  Decile 9 | 57.002 [46.279 to 68.773] | 118.576 [102.905 to 154.382]
  Decile 10: number analyzed (Participants) | 54 | 37
  Decile 10 | 95.573 [68.774 to 428.103] | 216.040 [154.383 to 1006.328]

16. Secondary Outcome: Comparison of Distribution of HPV18 Antibodies Levels Assessed at 24 Months
Description: Distribution of HPV18 antibodies levels assessed at 24 months following a single dose of Cervarix in 9-14 year old girls compared to distribution of HPV18 antibodies levels assessed at 24 months following three doses of Gardasil, administered at 0, 2, and 6 months, in 18-25 year old women. Shown as medians and ranges by deciles.
Time Frame: 24 months
Population: as for outcome 7
Measure: Median (Full Range); unit: International units (IU/mL)
Arm/Group | Girls (1D Cervarix®) | Women (3D Gardasil-4®)
Number analyzed (Participants) | 530 | 376
International units (IU/mL)
  Decile 1: number analyzed (Participants) | 53 | 38
  Decile 1 | 1.568 [0.520 to 2.169] | 1.563 [0.520 to 2.274]
  Decile 2: number analyzed (Participants) | 53 | 38
  Decile 2 | 2.757 [2.170 to 3.537] | 2.993 [2.275 to 3.661]
  Decile 3: number analyzed (Participants) | 53 | 37
  Decile 3 | 4.259 [3.538 to 4.876] | 4.118 [3.662 to 4.853]
  Decile 4: number analyzed (Participants) | 53 | 38
  Decile 4 | 5.465 [4.844 to 6.110] | 5.470 [4.854 to 6.465]
  Decile 5: number analyzed (Participants) | 53 | 37
  Decile 5 | 7.183 [6.111 to 8.105] | 7.759 [6.466 to 8.832]
  Decile 6: number analyzed (Participants) | 53 | 38
  Decile 6 | 9.274 [8.106 to 10.373] | 10.326 [8.833 to 11.590]
  Decile 7: number analyzed (Participants) | 53 | 38
  Decile 7 | 11.425 [10.374 to 13.536] | 12.739 [11.591 to 14.510]
  Decile 8: number analyzed (Participants) | 53 | 37
  Decile 8 | 15.207 [13.537 to 18.026] | 16.287 [14.511 to 20.471]
  Decile 9: number analyzed (Participants) | 53 | 38
  Decile 9 | 21.259 [18.027 to 28.251] | 26.680 [20.472 to 39.323]
  Decile 10: number analyzed (Participants) | 53 | 37
  Decile 10 | 39.083 [28.252 to 182.221] | 58.887 [39.324 to 264.857]

17. Secondary Outcome: Number Seropositive for HPV16 at 36 Months, Excluding 9-10 Year Olds
Description: Will measure HPV16 specific serum antibody using the HPV type-specific ELISA on serum. assessed at 36 months after initial vaccination, following a single dose of Cervarix in 11-14-year-old girls and three doses of Gardasil, administered at 0, 2, and 6 months, in 18-25 year old women. For computing proportions seropositive and proportions seroconverting, HPV16 is seropositive if the ELISA concentration is greater than 1.41 IU/mL. Participants whose analysis of the 36-month sample does not generate a valid HPV16 result will be excluded only from the 36-month HPV16 analysis.
Time Frame: 36 month
Population: The primary cohort for the analysis of HPV16 among girls 11-14 at and women at 36 months includes participants who received the appropriate number of vaccine doses within the specified windows, were initially seronegative for HPV16, underwent blood collection at the 36-month mark, and reported no additional HPV vaccinations outside the study before the 36-month blood collection, as confirmed by self-report or serologic testing for HPV6/HPV11.
Measure: Count of Participants; unit: Participants
Groups:
- 11-14-year-old Girls (1D Cervarix®): Participants 11-14 years old receive Cervarix IM at baseline. Recombinant Human Papillomavirus Bivalent Vaccine: Given IM
- Women (3D Gardasil-4®): Participants 18-25 years old receive Gardasil IM at baseline and at 2 and 6 months in the absence of unacceptable toxicity. Quadrivalent Human Papillomavirus (types 6, 11, 16, 18) Recombinant Vaccine: Given IM
Arm/Group | 11-14-year-old Girls (1D Cervarix®) | Women (3D Gardasil-4®)
Number analyzed (Participants) | 462 | 366
Participants | 461 | 366

18. Secondary Outcome: Comparison of GMCs for HPV16 Antibodies Assessed at 36 Months, Excluding 9-10-year-old Girls
Description: To compare GMCs for HPV16 antibodies, assessed at 36 months after initial vaccination, following a single dose of Cervarix in 11-14-year-old girls and three doses of Gardasil, administered at 0, 2, and 6 months, in 18-25 year old women.
Time Frame: 36 month
Population: as for outcome 17
Measure: Geometric Mean (95% Confidence Interval); unit: International units (IU/mL)
Groups:
- Girls (1D Cervarix®), Excluding 9-10 Year Old Girls: Participants 11-14 years old receive Cervarix IM at baseline.
Arm/Group | Girls (1D Cervarix®), Excluding 9-10 Year Old Girls | Women (3D Gardasil-4®)
Number analyzed (Participants) | 461 | 366
International units (IU/mL) | 20.8 [19.0 to 22.8] | 42.8 [38.8 to 47.2]
Statistical Analysis 1: Comparison: Girls (1D Cervarix®), Excluding 9-10 Year Old Girls vs Women (3D Gardasil-4®); Test type: Non-Inferiority — Let R=GMC1/GMC3 be the ratio of geometric mean concentrations of 1 dose to 3 doses. We reject the noninferiority hypothesis if at 36 months the lower limit of the two-sided 96% confidence interval on R ≥ 0.67 for HPV16 and HPV18. The overall Type 1 error rate for rejecting the null hypotheses for both HPV16 and HPV18 (i.e., declaring noninferiority of the 1D2V) at either time point was controlled at 0.025.); GMC Ratio = 0.49, 96% CI 2-sided [0.42 to 0.56] — Generalized estimating equations were used to estimate R and construct confidence intervals

19. Secondary Outcome: Comparison of Seroconversion Proportions for HPV16 Antibodies Assessed at 36 Months, Excluding 9-10-year-old Girls
Description: To compare seroconversion proportions for HPV16 antibodies, assessed at 36 months after initial vaccination, following a single dose of Cervarix in 11-14-year-old girls and three doses of Gardasil, administered at 0, 2, and 6 months, in 18-25 year old women.
Time Frame: 36 month
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Groups:
- Women (3D Gardasil®): Participants 18-25 years old receive Gardasil IM at baseline and at 2 and 6 months in the absence of unacceptable toxicity. Quadrivalent Human Papillomavirus (types 6, 11, 16, 18) Recombinant Vaccine: Given IM
Arm/Group | 11-14-year-old Girls (1D Cervarix®) | Women (3D Gardasil®)
Number analyzed (Participants) | 462 | 366
Participants | 461 | 366
Statistical Analysis 1: Comparison: 11-14-year-old Girls (1D Cervarix®) vs Women (3D Gardasil®); Test type: Equivalence — [test comment as in outcome 9, analysis 1]; p = 1.0, Fisher Exact

20. Secondary Outcome: Number Seropositive for HPV18 at 36 Months, Excluding 9-10 Year Olds
Description: Will measure HPV18 specific serum antibody using the HPV type-specific ELISA on serum. assessed at 36 months after initial vaccination, following a single dose of Cervarix in 11-14-year-old girls and three doses of Gardasil, administered at 0, 2, and 6 months, in 18-25 year old women. For computing proportions seropositive and proportions seroconverting, HPV18 is seropositive if the ELISA concentration is greater than 1.05 IU/mL. Participants whose analysis of the 36-month sample does not generate a valid HPV18 result will be excluded only from the 36-month HPV18 analysis.
Time Frame: 36 month
Population: The primary cohort for the analysis of HPV18 among girls 11-14 at and women at 36 months includes participants who received the appropriate number of vaccine doses within the specified windows, were initially seronegative for HPV18, underwent blood collection at the 36-month mark, and reported no additional HPV vaccinations outside the study before the 36-month blood collection, as confirmed by self-report or serologic testing for HPV6/HPV11.
Measure: Count of Participants; unit: Participants
Arm/Group | 11-14-year-old Girls (1D Cervarix®) | Women (3D Gardasil-4®)
Number analyzed (Participants) | 447 | 373
Participants | 441 | 358

21. Secondary Outcome: Comparison of GMCs for HPV18 Antibodies, Assessed at 36 Months, Excluding 9-10-year-old Girls
Description: To compare GMCs for HPV18 antibodies, assessed at 36 months after initial vaccination, following a single dose of Cervarix in 11-14-year-old girls and three doses of Gardasil, administered at 0, 2, and 6 months, in 18-25-year-old women.
Time Frame: 36 month
Population: as for outcome 20
Measure: Geometric Mean (95% Confidence Interval); unit: International units (IU/mL)
Arm/Group | Girls (1D Cervarix®), Excluding 9-10 Year Old Girls | Women (3D Gardasil-4®)
Number analyzed (Participants) | 441 | 358
International units (IU/mL) | 7.9 [7.2 to 8.7] | 7.2 [6.4 to 8.1]
Statistical Analysis 1: Comparison: Girls (1D Cervarix®), Excluding 9-10 Year Old Girls vs Women (3D Gardasil-4®); Test type: Non-Inferiority — [test comment as in outcome 18, analysis 1]; GMC Ratio = 1.09, 96% CI 2-sided [0.93 to 1.27]

22. Secondary Outcome: Comparison of Seroconversion Proportions for HPV18 Antibodies, Assessed at 36 Months, Excluding 9-10-year-old Girls
Description: To compare seroconversion proportions for HPV18 antibodies, assessed at 36 months after initial vaccination, following a single dose of Cervarix in 11-14-year-old girls and three doses of Gardasil, administered at 0, 2, and 6 months, in 18-25-year-old women.
Time Frame: 36 month
Population: The primary cohort for the analysis of HPV16 among girls 11-14 years old and women at 36 months includes participants who received the appropriate number of vaccine doses within the specified windows, were initially seronegative for HPV16, underwent blood collection at the 36-month mark, and reported no additional HPV vaccinations outside the study before the 36-month blood collection, as confirmed by self-report or serologic testing for HPV6/HPV11.
Measure: Count of Participants; unit: Participants
Arm/Group | Girls (1D Cervarix®), Excluding 9-10 Year Old Girls | Women (3D Gardasil-4®)
Number analyzed (Participants) | 447 | 373
Participants | 441 | 358
Statistical Analysis 1: Comparison: Girls (1D Cervarix®), Excluding 9-10 Year Old Girls vs Women (3D Gardasil-4®); Test type: Equivalence — [test comment as in outcome 9, analysis 1]; p = 0.0006, Fisher Exact

23. Secondary Outcome: Number Seropositive for HPV16 at 24 Months, Excluding 9-10 Year Olds
Description: Will measure HPV16 specific serum antibody using the HPV type-specific ELISA on serum. assessed at 24 months after initial vaccination, following a single dose of Cervarix in 11-14-year-old girls and three doses of Gardasil, administered at 0, 2, and 6 months, in 18-25 year old women. For computing proportions seropositive and proportions seroconverting, HPV16 is seropositive if the ELISA concentration is greater than 1.41 IU/mL. Participants whose analysis of the 24-month sample does not generate a valid HPV16 result will be excluded only from the 24-month HPV16 analysis.
Time Frame: 24 month
Population: The primary cohort for the analysis of HPV16 among girls 11-14 and women at 24 months includes participants who received the appropriate number of vaccine doses within the specified windows, were initially seronegative for HPV16, underwent blood collection at the 24-month mark, and reported no additional HPV vaccinations outside the study before the 24-month blood collection, as confirmed by self-report or serologic testing for HPV6/HPV11.
Measure: Count of Participants; unit: Participants
Arm/Group | 11-14-year-old Girls (1D Cervarix®) | Women (3D Gardasil-4®)
Number analyzed (Participants) | 464 | 371
Participants | 463 | 371

24. Secondary Outcome: Comparison of GMCs for HPV16 Assessed at 24 Months, Excluding 9-10-year-old Girls
Description: To compare GMCs for HPV16 antibodies, assessed at 24 months after initial vaccination, following a single dose of Cervarix in 11-14-year-old girls and three doses of Gardasil, administered at 0, 2, and 6 months, in 18-25-year-old women.
Time Frame: 24 months
Population: as for outcome 23
Measure: Geometric Mean (95% Confidence Interval); unit: International units (IU/mL)
Arm/Group | Girls (1D Cervarix®), Excluding 9-10 Year Old Girls | Women (3D Gardasil-4®)
Number analyzed (Participants) | 463 | 371
International units (IU/mL) | 20.0 [18.3 to 21.9] | 48.8 [44.4 to 53.7]
Statistical Analysis 1: Comparison: Girls (1D Cervarix®), Excluding 9-10 Year Old Girls vs Women (3D Gardasil-4®); Test type: Non-Inferiority — Let R=GMC1/GMC3 be the ratio of geometric mean concentrations of 1 dose to 3 doses. We reject the noninferiority hypothesis if at 24 months the lower limit of the two-sided 99% confidence interval on R ≥ 0.67 for HPV16 and HPV18. The overall Type 1 error rate for rejecting the null hypotheses for both HPV16 and HPV18 (i.e., declaring noninferiority of the 1D2V) at either time point was controlled at 0.025; GMC Ratio = 0.41, 99% CI 2-sided [0.35 to 0.49] — Generalized estimating equations were used to estimate R and construct confidence intervals

25. Secondary Outcome: Comparison of Seroconversion Proportions for HPV16 Assessed at 24 Months, Excluding 9-10-year-old Girls
Description: To compare seroconversion proportions for HPV16 antibodies, assessed at 24 months after initial vaccination, following a single dose of Cervarix in 11-14-year-old girls and three doses of Gardasil, administered at 0, 2, and 6 months, in 18-25-year-old women.
Time Frame: 24 months
Population: The primary cohort for the interim analysis of HPV16 includes 11-14-year-old girls and women who received the appropriate number of vaccine doses within the specified windows, were initially seronegative for HPV16, underwent blood collection at the 24-month mark, and reported no additional HPV vaccinations outside the study before the 24-month blood collection, as confirmed by self-report or serologic testing for HPV6/HPV11.
Measure: Count of Participants; unit: Participants
Groups:
- 11-14 Year Old Girls (1D Cervarix®): Participants 11-14 years old receive Cervarix IM at baseline. Recombinant Human Papillomavirus Bivalent Vaccine: Given IM
Arm/Group | 11-14 Year Old Girls (1D Cervarix®) | Women (3D Gardasil-4®)
Number analyzed (Participants) | 464 | 371
Participants | 463 | 371
Statistical Analysis 1: Comparison: 11-14 Year Old Girls (1D Cervarix®) vs Women (3D Gardasil-4®); Test type: Equivalence — [test comment as in outcome 9, analysis 1]; p = 1.0, Fisher Exact

26. Secondary Outcome: Number Seropositive for HPV18 at 24 Months, Excluding 9-10 Year Olds
Description: Will measure HPV18 specific serum antibody using the HPV type-specific ELISA on serum. assessed at 24 months after initial vaccination, following a single dose of Cervarix in 11-14-year-old girls and three doses of Gardasil, administered at 0, 2, and 6 months, in 18-25 year old women. For computing proportions seropositive and proportions seroconverting, HPV18 is seropositive if the ELISA concentration is greater than 1.05 IU/mL. Participants whose analysis of the 24-month sample does not generate a valid HPV18 result will be excluded only from the 24-month HPV18 analysis.
Time Frame: 24 month
Population: The primary cohort for the interim analysis of HPV18 includes 11-14-year-old girls and women who received the appropriate number of vaccine doses within the specified windows, were initially seronegative for HPV18, underwent blood collection at the 24-month mark, and reported no additional HPV vaccinations outside the study before the 24-month blood collection, as confirmed by self-report or serologic testing for HPV6/HPV11.
Measure: Count of Participants; unit: Participants
Arm/Group | 11-14-year-old Girls (1D Cervarix®) | Women (3D Gardasil-4®)
Number analyzed (Participants) | 448 | 376
Participants | 440 | 367

27. Secondary Outcome: Comparison of GMCs for HPV18 Antibodies, Assessed at 24 Months, Excluding 9-10-year-old Girls
Description: To compare GMCs for HPV18 antibodies, assessed at 24 months after initial vaccination, following a single dose of Cervarix in 11-14-year-old girls and three doses of Gardasil, administered at 0, 2, and 6 months, in 18-25-year-old women.
Time Frame: 24 months
Measure: Geometric Mean (95% Confidence Interval); unit: International units (IU/mL)
Arm/Group | 11-14-year-old Girls (1D Cervarix®) | Women (3D Gardasil-4®)
Number analyzed (Participants) | 440 | 367
International units (IU/mL) | 7.6 [6.9 to 8.3] | 8.8 [7.9 to 9.9]
Statistical Analysis 1: Comparison: 11-14-year-old Girls (1D Cervarix®) vs Women (3D Gardasil-4®); Test type: Non-Inferiority — [test comment as in outcome 24, analysis 1]; GMC Ratio = 0.86, 99% CI 2-sided [0.71 to 1.04] — Generalized estimating equations were used to estimate R and construct confidence intervals

28. Secondary Outcome: Comparison of Seroconversion Proportions for HPV18 Antibodies, Assessed at 24 Months, Excluding 9-10-year-old Girls
Description: To compare seroconversion proportions for HPV18 antibodies, assessed at 24 months after initial vaccination, following a single dose of Cervarix in 11-14-year-old girls and three doses of Gardasil, administered at 0, 2, and 6 months, in 18-25-year-old women.
Time Frame: 24 months
Population: The cohort for this analysis at 24 months includes girls 11-14 and women who received the appropriate number of vaccine doses within the specified windows, were initially seronegative for HPV18, underwent blood collection at the 24-month mark, and reported no additional HPV vaccinations outside the study before the 24-month blood collection, as confirmed by self-report or serologic testing for HPV6/HPV11.
Measure: Count of Participants; unit: Participants
Arm/Group | 11-14-year-old Girls (1D Cervarix®) | Women (3D Gardasil-4®)
Number analyzed (Participants) | 448 | 376
Participants | 440 | 367
Statistical Analysis 1: Comparison: 11-14-year-old Girls (1D Cervarix®) vs Women (3D Gardasil-4®); Test type: Equivalence — [test comment as in outcome 9, analysis 1]; p = 0.478, Fisher Exact

29. Secondary Outcome: Number Seropositive for HPV16 Antibodies, Assessed at 1 Month After Vaccination, in Younger and Older Girls
Description: Will measure HPV16 specific serum antibody using the HPV type-specific ELISA on serum. For computing proportions seropositive and proportions seroconverting, HPV16 is seropositive if the ELISA titer is greater than 1.41 IU/mL. Participants whose analysis of the 1-month sample does not generate a valid HPV16 result will be excluded only from the 1-month HPV16 analysis.
Time Frame: 1 month
Population: The cohort for the 1 month analysis of HPV16 includes 9-14 year old girls who received the appropriate number of vaccine doses within the specified windows, were initially seronegative for HPV16, underwent blood collection at the 1-month mark, and reported no additional HPV vaccinations outside the study before the 1-month blood collection, as confirmed by self-report or serologic testing for HPV6/HPV11.
Measure: Count of Participants; unit: Participants
Groups:
- 9-10 Years Old Girls (1D Cervarix®): Participants 9-10 years old receive Cervarix IM at baseline. Recombinant Human Papillomavirus Bivalent Vaccine: Given IM
Arm/Group | 9-10 Years Old Girls (1D Cervarix®) | 11-14-year-old Girls (1D Cervarix®)
Number analyzed (Participants) | 99 | 461
Participants | 99 | 461

30. Secondary Outcome: Comparison of GMCs for HPV16 Antibodies, Assessed at 1 Month After Vaccination in Younger and Older Girls
Description: To compare GMCs for HPV16 antibodies, assessed at 1 month after vaccination, following a single dose of Cervarix in 9-10-year-old girls and following a single dose of Cervarix in 11-14-year-old girls, in order to compare girls who were in and not in the age range for routine HPV vaccination in Costa Rica.
Time Frame: 1 month
Population: as for outcome 29
Measure: Geometric Mean (95% Confidence Interval); unit: International units (IU/mL)
Groups:
- 9-10-year-old Girls (1D Cervarix®): Participants 9-10 years old receive Cervarix IM at baseline. Recombinant Human Papillomavirus Bivalent Vaccine: Given IM
Arm/Group | 9-10-year-old Girls (1D Cervarix®) | 11-14-year-old Girls (1D Cervarix®)
Number analyzed (Participants) | 99 | 461
International units (IU/mL) | 83.4 [71.2 to 97.8] | 62.6 [58.3 to 67.3]
Statistical Analysis 1: Comparison: 9-10-year-old Girls (1D Cervarix®) vs 11-14-year-old Girls (1D Cervarix®); Test type: Non-Inferiority — We reject the noninferiority hypothesis if the lower limit of the two-sided 95% confidence interval on R ≥ 0.67 for HPV16 and HPV18; GMC Ratio = 1.33, 95% CI 2-sided [1.12 to 1.58] — Generalized estimating equations were used to estimate R and construct confidence intervals

31. Secondary Outcome: Comparison of Seroconversion Proportions for HPV16 Antibodies, Assessed at 1 Month After Vaccination in Younger and Older Girls
Description: To compare seroconversion proportions for HPV16 antibodies, assessed at 1 month after vaccination, following a single dose of Cervarix in 9-10-year-old girls and following a single dose of Cervarix in 11-14-year-old girls.
Time Frame: 1 month
Population: Since both groups had a 100% seroconversion proportion, p-value could not be calculated.
Measure: Count of Participants; unit: Participants
Groups:
- 9-10 Year Old Girls (1D Cervarix®): Participants 9-10 years old receive Cervarix IM at baseline. Recombinant Human Papillomavirus Bivalent Vaccine: Given IM
Arm/Group | 9-10 Year Old Girls (1D Cervarix®) | 11-14-year-old Girls (1D Cervarix®)
Number analyzed (Participants) | 99 | 461
Participants | 99 | 461

32. Secondary Outcome: Number Seropositive for HPV18 Antibodies, Assessed at 1 Month After Vaccination, in Younger and Older Girls
Description: Will measure HPV18 specific serum antibody using the HPV type-specific ELISA on serum. For computing proportions seropositive and proportions seroconverting, HPV18 is seropositive if the ELISA titer is greater than 1.05 IU/mL. Participants whose analysis of the 1-month sample does not generate a valid HPV18 result will be excluded only from the 1-month HPV18 analysis.
Time Frame: 1 month
Population: The primary cohort for the 1-month analysis of HPV18 includes girls who received the appropriate number of vaccine doses within the specified windows, were initially seronegative for HPV18, underwent blood collection at the 1-month mark, and reported no additional HPV vaccinations outside the study before the 24-month blood collection, as confirmed by self-report or serologic testing for HPV6/HPV11.
Measure: Count of Participants; unit: Participants
Arm/Group | 9-10 Years Old Girls (1D Cervarix®) | 11-14-year-old Girls (1D Cervarix®)
Number analyzed (Participants) | 100 | 446
Participants | 100 | 446

33. Secondary Outcome: Comparison of GMCs for HPV18 Antibodies, Assessed at 1 Month After Vaccination in Younger and Older Girls
Description: To compare seroconversion proportions for HPV18 antibodies, assessed at 1 month after vaccination, following a single dose of Cervarix in 9-10-year-old girls and following a single dose of Cervarix in 11-14-year-old girls, in order to compare girls who were in and not in the age range for routine HPV vaccination in Costa Rica.
Time Frame: 1 month
Population: The primary cohort for the analysis of HPV18 among girls 9-14 at 1 month includes participants who received the appropriate number of vaccine doses within the specified windows, were initially seronegative for HPV18, underwent blood collection at the 1-month mark, and reported no additional HPV vaccinations outside the study before the 1-month blood collection, as confirmed by self-report or serologic testing for HPV6/HPV11.
Measure: Geometric Mean (95% Confidence Interval); unit: International units (IU/mL)
Arm/Group | 9-10 Year Old Girls (1D Cervarix®) | 11-14 Year Old Girls (1D Cervarix®)
Number analyzed (Participants) | 100 | 446
International units (IU/mL) | 32.8 [28.2 to 38.2] | 25.4 [23.3 to 27.6]
Statistical Analysis 1: Comparison: 9-10 Year Old Girls (1D Cervarix®) vs 11-14 Year Old Girls (1D Cervarix®); Test type: Non-Inferiority — [test comment as in outcome 30, analysis 1]; GMC Ratio = 1.29, 95% CI 2-sided [1.09 to 1.54] — Generalized estimating equations were used to estimate R and construct confidence intervals

34. Secondary Outcome: Comparison of Seroconversion Proportions for HPV18 Antibodies, Assessed at 1 Month After Vaccination in Younger and Older Girls
Description: as for outcome 33
Time Frame: 1 month
Population: Since both groups had a 100% seroconversion proportion, p-value could not be calculated.
Measure: Count of Participants; unit: Participants
Arm/Group | 9-10-year-old Girls (1D Cervarix®) | 11-14-year-old Girls (1D Cervarix®)
Number analyzed (Participants) | 100 | 446
Participants | 100 | 446

35. Secondary Outcome: Number Seropositive for HPV16 Antibodies, Assessed at 12 Months After Vaccination, in Younger and Older Girls
Description: Will measure HPV16 specific serum antibody using the HPV type-specific ELISA on serum. For computing proportions seropositive and proportions seroconverting, HPV16 is seropositive if the ELISA titer is greater than 1.41 IU/mL. Participants whose analysis of the 12-month sample does not generate a valid HPV16 result will be excluded only from the 12-month HPV16 analysis.
Time Frame: 12 months
Population: The cohort for the 12-month analysis of HPV16 includes girls 9-14 years old who received the appropriate number of vaccine doses within the specified windows, were initially seronegative for HPV16, underwent blood collection at the 12-month mark, and reported no additional HPV vaccinations outside the study before the 12-month blood collection, as confirmed by self-report or serologic testing for HPV6/HPV11.
Measure: Count of Participants; unit: Participants
Arm/Group | 9-10 Years Old Girls (1D Cervarix®) | 11-14-year-old Girls (1D Cervarix®)
Number analyzed (Participants) | 85 | 464
Participants | 85 | 462

36. Secondary Outcome: Comparison of GMCs for HPV16 Antibodies, Assessed at 12 Months After Vaccination in Younger and Older Girls
Description: To compare GMCs for HPV16 antibodies, assessed at 12 months after vaccination, following a single dose of Cervarix in 9-10-year-old girls and following a single dose of Cervarix in 11-14-year-old girls, in order to compare girls who were in and not in the age range for routine HPV vaccination in Costa Rica.
Time Frame: 1 year
Population: The cohort for the analysis of HPV16 at 12 months includes girls 9-14 years old who received the appropriate number of vaccine doses within the specified windows, were initially seronegative for HPV16, underwent blood collection at the 12-month mark, and reported no additional HPV vaccinations outside the study before the 12-month blood collection, as confirmed by self-report or serologic testing for HPV6/HPV11.
Measure: Geometric Mean (95% Confidence Interval); unit: International units (IU/mL)
Arm/Group | 9-10-year-old Girls (1D Cervarix®) | 11-14-year-old Girls (1D Cervarix®)
Number analyzed (Participants) | 85 | 462
International units (IU/mL) | 25.0 [20.7 to 30.2] | 17.0 [15.5 to 18.6]
Statistical Analysis 1: Comparison: 9-10-year-old Girls (1D Cervarix®) vs 11-14-year-old Girls (1D Cervarix®); Test type: Non-Inferiority — [test comment as in outcome 30, analysis 1]; GMC Ratio = 1.48, 95% CI 2-sided [1.20 to 1.81] — Generalized estimating equations were used to estimate R and construct confidence intervals

37. Secondary Outcome: Comparison of Seroconversion Proportions for HPV16 Antibodies, Assessed at 12 Months After Vaccination in Younger and Older Girls
Description: To compare seroconversion proportions for HPV16 antibodies, assessed at 12 months after vaccination, following a single dose of Cervarix in 9-10-year-old girls and following a single dose of Cervarix in 11-14-year-old girls.
Time Frame: 1 year
Population: as for outcome 36
Measure: Count of Participants; unit: Participants
Arm/Group | 9-10 Year Old Girls (1D Cervarix®) | 11-14-year-old Girls (1D Cervarix®)
Number analyzed (Participants) | 85 | 464
Participants | 85 | 462
Statistical Analysis 1: Comparison: 9-10 Year Old Girls (1D Cervarix®) vs 11-14-year-old Girls (1D Cervarix®); Test type: Equivalence — We will use a Fisher Exact test to test for the difference of the seroconversion rate between one-dose 9-10 year old girls and one-dose 11-14 year old girls. A p-value under 0.05 will be regarded as significant; p = 1.0, Fisher Exact

38. Secondary Outcome: Number Seropositive for HPV18 Antibodies, Assessed at 12 Months After Vaccination, in Younger and Older Girls
Description: Will measure HPV18 specific serum antibody using the HPV type-specific ELISA on serum. For computing proportions seropositive and proportions seroconverting, HPV18 is seropositive if the ELISA titer is greater than 1.05 IU/mL. Participants whose analysis of the 12-month sample does not generate a valid HPV18 result will be excluded only from the 12-month HPV18 analysis.
Time Frame: 12 month
Population: The primary cohort for the 12-month analysis of HPV18 includes 9-14 year old girls who received the appropriate number of vaccine doses within the specified windows, were initially seronegative for HPV18, underwent blood collection at the 12-month mark, and reported no additional HPV vaccinations outside the study before the 12-month blood collection.
Measure: Count of Participants; unit: Participants
Arm/Group | 9-10 Years Old Girls (1D Cervarix®) | 11-14-year-old Girls (1D Cervarix®)
Number analyzed (Participants) | 84 | 448
Participants | 84 | 440

39. Secondary Outcome: Comparison of GMCs for HPV18 Antibodies, Assessed at 12 Months After Vaccination in Younger and Older Girls
Description: To compare GMCs for HPV18 antibodies, assessed at 12 months after vaccination, following a single dose of Cervarix in 9-10-year-old girls and following a single dose of Cervarix in 11-14-year-old girls. in order to compare girls who were in and not in the age range for routine HPV vaccination in Costa Rica.
Time Frame: 12 months
Population: The cohort for the analysis of HPV18 at 12 months includes girls 9-14 years old who received the appropriate number of vaccine doses within the specified windows, were initially seronegative for HPV18, underwent blood collection at the 12-month mark, and reported no additional HPV vaccinations outside the study before the 12-month blood collection, as confirmed by self-report or serologic testing for HPV6/HPV11.
Measure: Geometric Mean (95% Confidence Interval); unit: International units (IU/mL)
Arm/Group | 9-10-year-old Girls (1D Cervarix®) | 11-14-year-old Girls (1D Cervarix®)
Number analyzed (Participants) | 84 | 440
International units (IU/mL) | 10.6 [8.8 to 12.9] | 7.5 [6.9 to 8.2]
Statistical Analysis 1: Comparison: 9-10-year-old Girls (1D Cervarix®) vs 11-14-year-old Girls (1D Cervarix®); Test type: Non-Inferiority — [test comment as in outcome 30, analysis 1]; GMC Ratio = 1.42, 95% CI 2-sided [1.15 to 1.75] — Generalized estimating equations were used to estimate R and construct confidence intervals

40. Secondary Outcome: Comparison of Seroconversion Proportions for HPV18 Antibodies, Assessed at 12 Months After Vaccination, in Younger and Older Girls
Description: To compare seroconversion proportions for HPV18 antibodies, assessed at 1 year after vaccination, following a single dose of Cervarix in 9-10-year-old girls and following a single dose of Cervarix in 11-14-year-old girls, in order to compare girls who were in and not in the age range for routine HPV vaccination in Costa Rica.
Time Frame: 1 year
Population: as for outcome 39
Measure: Count of Participants; unit: Participants
Arm/Group | 9-10-year-old Girls (1D Cervarix®) | 11-14-year-old Girls (1D Cervarix®)
Number analyzed (Participants) | 84 | 448
Participants | 84 | 440
Statistical Analysis 1: Comparison: 9-10-year-old Girls (1D Cervarix®) vs 11-14-year-old Girls (1D Cervarix®); Test type: Equivalence — [test comment as in outcome 37, analysis 1]; p = 0.368, Fisher Exact

41. Secondary Outcome: Number Seropositive for HPV16 at 36 Months, By Enrollment Age Group
Description: Will measure HPV16 specific serum antibody using the HPV type-specific ELISA on serum. For computing proportions seropositive and proportions seroconverting, HPV16 is seropositive if the ELISA titer is greater than 1.41 IU/mL. Participants whose analysis of the 36-month sample does not generate a valid HPV16 result will be excluded only from the 36-month HPV16 analysis.
Time Frame: 36 months
Population: The primary cohort for the analysis of HPV16 by enrollment age grouping includes participants who received the appropriate number of vaccine doses within the specified windows, were initially seronegative for HPV16, underwent blood collection at the 36-month mark, and reported no additional HPV vaccinations outside the study before the 36-month blood collection, as confirmed by self-report or serologic testing for HPV6/HPV11
Measure: Count of Participants; unit: Participants
Groups:
- 9-11 Year Old Girls (1D Cervarix®): Participants 9-11 years old receive Cervarix IM at baseline. Recombinant Human Papillomavirus Bivalent Vaccine: Given IM
- 12-14-year-old Girls (1D Cervarix®): Participants 12-14 years old receive Cervarix IM at baseline. Recombinant Human Papillomavirus Bivalent Vaccine: Given IM
- 18-21 Year Old Women (3D Gardasil-4®): Participants 18-21 years old receive Gardasil IM at baseline and at 2 and 6 months in the absence of unacceptable toxicity. Quadrivalent Human Papillomavirus (types 6, 11, 16, 18) Recombinant Vaccine: Given IM
- 22-25 Year Old Women (3D Gardasil-4®): Participants 22-25 years old receive Gardasil IM at baseline and at 2 and 6 months in the absence of unacceptable toxicity. Quadrivalent Human Papillomavirus (types 6, 11, 16, 18) Recombinant Vaccine: Given IM
Arm/Group | 9-11 Year Old Girls (1D Cervarix®) | 12-14-year-old Girls (1D Cervarix®) | 18-21 Year Old Women (3D Gardasil-4®) | 22-25 Year Old Women (3D Gardasil-4®)
Number analyzed (Participants) | 203 | 336 | 226 | 140
Participants | 203 | 335 | 226 | 140

42. Secondary Outcome: Comparison of GMCs for HPV16 Antibodies Assessed at 36 Months, by Enrollment Age Group
Description: To evaluate whether age is associated with GMCs for HPV16 antibodies, assessed at 36 months after initial vaccination.
Time Frame: 36 month
Population: The cohort for the analysis of HPV16 at 36 months by enrollment age group includes participants who received the appropriate number of vaccine doses within the specified windows, were initially seronegative for HPV16, underwent blood collection at the 36-month mark, and reported no additional HPV vaccinations outside the study before the 36-month blood collection, as confirmed by self-report or serologic testing for HPV6/HPV11.
Measure: Geometric Mean (95% Confidence Interval); unit: International units (IU/mL)
Groups:
- 22-25 Year Old Women (3D Gardasil-4®): Participants 18-25 years old receive Gardasil IM at baseline and at 2 and 6 months in the absence of unacceptable toxicity. Quadrivalent Human Papillomavirus (types 6, 11, 16, 18) Recombinant Vaccine: Given IM
Arm/Group | 9-11 Year Old Girls (1D Cervarix®) | 12-14-year-old Girls (1D Cervarix®) | 18-21 Year Old Women (3D Gardasil-4®) | 22-25 Year Old Women (3D Gardasil-4®)
Number analyzed (Participants) | 203 | 335 | 226 | 140
International units (IU/mL) | 21.7 [19.1 to 24.6] | 21.2 [19.0 to 23.6] | 47.1 [41.5 to 53.4] | 36.7 [31.7 to 42.5]
Statistical Analysis 1: Comparison: 9-11 Year Old Girls (1D Cervarix®) vs 18-21 Year Old Women (3D Gardasil-4®); This procedure controls the overall type one error at 0.05. We are conducting 4 one-sided tests and will spend alpha as follows: 0.005 of the alpha each for HPV16 and for HPV18 at 24 months and 0.02 of the alpha each for HPV16 and for HPV18 at 36 months. The experiment-wise significance level accounting for multiple comparisons is ≤0.05 because the null chance of rejection for either HPV16or HPV18 is ≤0.01 at 24 months by the Bonferroni inequality and ≤0.04 at 36 months; Test type: Non-Inferiority — [test comment as in outcome 18, analysis 1]; GMC Ratio = 0.46, 96% CI 2-sided [0.38 to 0.56] — Generalized estimating equations were used to estimate R and construct confidence intervals
Statistical Analysis 2: Comparison: 12-14-year-old Girls (1D Cervarix®) vs 22-25 Year Old Women (3D Gardasil-4®); Test type: Non-Inferiority — [test comment as in outcome 18, analysis 1]; GMC Ratio = .58, 96% CI 2-sided [0.48 to 0.70] — Generalized estimating equations were used to estimate R and construct confidence intervals
Statistical Analysis 3: Comparison: 9-11 Year Old Girls (1D Cervarix®) vs 12-14-year-old Girls (1D Cervarix®) vs 18-21 Year Old Women (3D Gardasil-4®) vs 22-25 Year Old Women (3D Gardasil-4®); Test type: Equivalence — A p-value <0.05 is interpreted as significantly different GMC ratios in different strata; p = 0.079, p-values test for heterogeneity — The p-values test for heterogeneity in the GMC ratios estimated from the stratified analyses

43. Secondary Outcome: Comparison of Seroconversion Proportions for HPV16, Assessed at 36 Months, by Enrollment Age Group
Description: To evaluate whether age is associated with seroconversion proportions for HPV-16 antibodies, assessed at 36 months after initial vaccination.
Time Frame: 36 month
Measure: Count of Participants; unit: Participants
Groups:
- 18-21 Year Old Women (3D Gardasil-4®): Participants 18-25 years old receive Gardasil IM at baseline and at 2 and 6 months in the absence of unacceptable toxicity. Quadrivalent Human Papillomavirus (types 6, 11, 16, 18) Recombinant Vaccine: Given IM
Arm/Group | 9-11 Year Old Girls (1D Cervarix®) | 12-14-year-old Girls (1D Cervarix®) | 18-21 Year Old Women (3D Gardasil-4®) | 22-25 Year Old Women (3D Gardasil-4®)
Number analyzed (Participants) | 203 | 336 | 226 | 140
Participants | 203 | 335 | 226 | 140
Statistical Analysis 1: Comparison: 12-14-year-old Girls (1D Cervarix®) vs 22-25 Year Old Women (3D Gardasil-4®); NOTE: Younger one-dose recipients (9-11 Year Old Girls) and three-dose recipients (18-21 Year Old Women) both had a 100% seroconversion proportion for HPV16 at 36 months, so a p-value for the difference of the seroconversion rate between them could not be calculated. Therefore, we only include the calculated p-value for the comparison of the seroconversion rate between older one-dose recipients (9-11 Year Old Girls) and three-dose recipients (22-25 Year Old Women); Test type: Equivalence — We will use a Fisher Exact test to test for the difference of the seroconversion rate between the older one-dose recipients and the older three-dose recipients. A p-value under 0.05 will be regarded as significant; p = 1.0000, Fisher Exact

44. Secondary Outcome: Number Seropositive for HPV18 at 36 Months, By Enrollment Age Group
Description: Will measure HPV18 specific serum antibody using the HPV type-specific ELISA on serum. For computing proportions seropositive and proportions seroconverting, HPV18 is seropositive if the ELISA titer is greater than 1.05 IU/mL. Participants whose analysis of the 36-month sample does not generate a valid HPV18 result will be excluded only from the 36-month HPV18 analysis.
Time Frame: 36 months
Population: The primary cohort for the analysis of HPV18 by enrollment age group includes participants who received the appropriate number of vaccine doses within the specified windows, were initially seronegative for HPV18, underwent blood collection at the 36-month mark, and reported no additional HPV vaccinations outside the study before the 36-month blood collection, as confirmed by self-report or serologic testing for HPV6/HPV11.
Measure: Count of Participants; unit: Participants
Arm/Group | 9-11 Year Old Girls (1D Cervarix®) | 12-14-year-old Girls (1D Cervarix®) | 18-21 Year Old Women (3D Gardasil-4®) | 22-25 Year Old Women (3D Gardasil-4®)
Number analyzed (Participants) | 199 | 324 | 212 | 161
Participants | 199 | 318 | 201 | 157

45. Secondary Outcome: Comparison of GMCs for HPV18 Antibodies, Assessed at 36 Months, by Enrollment Age Group
Description: To evaluate whether age is associated with GMCs for HPV18 antibodies, assessed at 36 months after initial vaccination.
Time Frame: 36 month
Population: The cohort for the analysis of HPV18 at 36 months by enrollment age group includes participants who received the appropriate number of vaccine doses within the specified windows, were initially seronegative for HPV18, underwent blood collection at the 36-month mark, and reported no additional HPV vaccinations outside the study before the 36-month blood collection, as confirmed by self-report or serologic testing for HPV6/HPV11.
Measure: Geometric Mean (95% Confidence Interval); unit: International units (IU/mL)
Groups:
- 9-11 Girls (1D Cervarix): Participants 9-11 years old receive Cervarix IM at baseline. Recombinant Human Papillomavirus Bivalent Vaccine: Given IM
- 12-14 Girls (1D Cervarix): Participants 12-14 years old receive Cervarix IM at baseline. Recombinant Human Papillomavirus Bivalent Vaccine: Given IM
- 18-21 Women (3D Gardasil): Participants 18-21 years old receive Gardasil IM at baseline and at 2 and 6 months in the absence of unacceptable toxicity. Quadrivalent Human Papillomavirus (types 6, 11, 16, 18) Recombinant Vaccine: Given IM
- 22-25 Women (3D Gardasil): Participants 22-25 years old receive Gardasil IM at baseline and at 2 and 6 months in the absence of unacceptable toxicity. Quadrivalent Human Papillomavirus (types 6, 11, 16, 18) Recombinant Vaccine: Given IM
Arm/Group | 9-11 Girls (1D Cervarix) | 12-14 Girls (1D Cervarix) | 18-21 Women (3D Gardasil) | 22-25 Women (3D Gardasil)
Number analyzed (Participants) | 199 | 318 | 201 | 157
International units (IU/mL) | 8.1 [7.2 to 9.2] | 7.9 [7.1 to 8.9] | 8.0 [6.8 to 9.5] | 6.4 [5.4 to 7.5]
Statistical Analysis 1: Comparison: 9-11 Girls (1D Cervarix) vs 18-21 Women (3D Gardasil); [analysis description as in outcome 42, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 18, analysis 1]; GMC Ratio = 1.01, 96% CI 2-sided [0.82 to 1.25]
Statistical Analysis 2: Comparison: 12-14 Girls (1D Cervarix) vs 22-25 Women (3D Gardasil); The cohort for the analysis of HPV16 at 36 months by enrollment age group includes participants who received the appropriate number of vaccine doses within the specified windows, were initially seronegative for HPV16, underwent blood collection at the 36-month mark, and reported no additional HPV vaccinations outside the study before the 36-month blood collection, as confirmed by self-report or serologic testing for HPV6/HPV11; Test type: Non-Inferiority — [test comment as in outcome 18, analysis 1]; GMC Ratio = 1.24, 96% CI 2-sided [1.01 to 1.54]
Statistical Analysis 3: Comparison: 9-11 Girls (1D Cervarix) vs 12-14 Girls (1D Cervarix) vs 18-21 Women (3D Gardasil) vs 22-25 Women (3D Gardasil); Test type: Equivalence — A p-value <0.05 is interpreted as significantly different GMC ratios in different strata; p = 0.14, p-values test for heterogeneity — The p-values test for heterogeneity in the GMC ratios estimated from the stratified analyses

46. Secondary Outcome: Comparison of Seroconversion Proportions for HPV18, Assessed at 36 Months, by Enrollment Age Group
Description: as for outcome 43
Time Frame: 36 month
Population: as for outcome 45
Measure: Count of Participants; unit: Participants
Groups:
- 9-11 Girls (1D Cervarix); 12-14 Girls (1D Cervarix): Participants 9-14 years old receive Cervarix IM at baseline. Recombinant Human Papillomavirus Bivalent Vaccine: Given IM
- 18-21 Women (3D Gardasil): Participants 18-25 years old receive Gardasil IM at baseline and at 2 and 6 months in the absence of unacceptable toxicity. Quadrivalent Human Papillomavirus (types 6, 11, 16, 18) Recombinant Vaccine: Given IM
Arm/Group | 9-11 Girls (1D Cervarix) | 12-14 Girls (1D Cervarix) | 18-21 Women (3D Gardasil) | 22-25 Women (3D Gardasil)
Number analyzed (Participants) | 199 | 324 | 212 | 161
Participants | 199 | 318 | 201 | 157
Statistical Analysis 1: Comparison: 9-11 Girls (1D Cervarix) vs 18-21 Women (3D Gardasil); Calculated p-value for the comparison of the seroconversion rate for HPV18 at 36 months between younger one-dose recipients (9-11 Year Old Girls) and the younger three-dose recipients (18-21 Year Old Women); Test type: Equivalence — We will use a Fisher Exact test to test for the difference of the seroconversion rate between the younger one-dose recipients and the younger three-dose recipients; p = 0.001, Fisher Exact — A p-value under 0.05 will be regarded as significant
Statistical Analysis 2: Comparison: 12-14 Girls (1D Cervarix) vs 22-25 Women (3D Gardasil); Calculated p-value for the comparison of the seroconversion rate for HPV18 at 36 months between older one-dose recipients (12-14 Year Old Girls) and the older three-dose recipients (22-25 Year Old Women); Test type: Equivalence — We will use a Fisher Exact test to test for the difference of the seroconversion rate between older one-dose and older three-dose recipients. A p-value under 0.05 will be regarded as significant; p = 0.737, Fisher Exact — A p-value under 0.05 will be regarded as significant

47. Secondary Outcome: Number Seropositive for HPV16 at 24 Months, By Enrollment Age Group
Description: as for outcome 5
Time Frame: 36 months
Population: The cohort for the analysis of HPV16 at 24 months by enrollment age grouping includes participants who received the appropriate number of vaccine doses within the specified windows, were initially seronegative for HPV16, underwent blood collection at the 24-month mark, and reported no additional HPV vaccinations outside the study before the 24-month blood collection, as confirmed by self-report or serologic testing for HPV6/HPV11
Measure: Count of Participants; unit: Participants
Arm/Group | 9-11 Year Old Girls (1D Cervarix®) | 12-14-year-old Girls (1D Cervarix®) | 18-21 Year Old Women (3D Gardasil-4®) | 22-25 Year Old Women (3D Gardasil-4®)
Number analyzed (Participants) | 211 | 336 | 229 | 142
Participants | 211 | 335 | 229 | 142

48. Secondary Outcome: Comparison of GMCs for HPV16 Antibodies Assessed at 24 Months, by Enrollment Age Group
Description: To evaluate whether age is associated with GMCs for HPV16 antibodies, assessed at 24 months after initial vaccination.
Time Frame: 24 month
Population: The cohort for the analysis of HPV16 at 24 months by enrollment age group includes participants who received the appropriate number of vaccine doses within the specified windows, were initially seronegative for HPV16, underwent blood collection at the 24-month mark, and reported no additional HPV vaccinations outside the study before the 24-month blood collection, as confirmed by self-report or serologic testing for HPV6/HPV11.
Measure: Geometric Mean (95% Confidence Interval); unit: International units (IU/mL)
Arm/Group | 9-11 Year Old Girls (1D Cervarix®) | 12-14-year-old Girls (1D Cervarix®) | 18-21 Year Old Women (3D Gardasil-4®) | 22-25 Year Old Women (3D Gardasil-4®)
Number analyzed (Participants) | 211 | 335 | 229 | 142
International units (IU/mL) | 22.0 [19.3 to 25.0] | 19.8 [17.8 to 22.0] | 53.2 [47.1 to 60.1] | 42.0 [36.2 to 48.7]
Statistical Analysis 1: Comparison: 9-11 Year Old Girls (1D Cervarix®) vs 18-21 Year Old Women (3D Gardasil-4®); [analysis description as in outcome 42, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 24, analysis 1]; GMC Ratio = 0.41, 99% CI 2-sided [0.33 to 0.52]
Statistical Analysis 2: Comparison: 12-14-year-old Girls (1D Cervarix®) vs 22-25 Year Old Women (3D Gardasil-4®); [analysis description as in outcome 42, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 24, analysis 1]; GMC Ratio = 0.47, 99% CI 2-sided [0.37 to 0.60]
Statistical Analysis 3: Comparison: 9-11 Year Old Girls (1D Cervarix®) vs 12-14-year-old Girls (1D Cervarix®) vs 18-21 Year Old Women (3D Gardasil-4®) vs 22-25 Year Old Women (3D Gardasil-4®); Test type: Equivalence — The p-values test for heterogeneity in the GMC ratios estimated from the stratified analyses; p = 0.028, p-values test for heterogeneity — A p-value <0.05 is interpreted as significantly different GMC ratios in different strata

49. Secondary Outcome: Comparison of Seroconversion Proportions for HPV16, Assessed at 24 Months, by Enrollment Age Group
Description: To evaluate whether age is associated with seroconversion proportions for HPV-16 antibodies, assessed at 24 months after initial vaccination.
Time Frame: 24 month
Population: as for outcome 48
Measure: Count of Participants; unit: Participants
Arm/Group | 9-11 Year Old Girls (1D Cervarix®) | 12-14-year-old Girls (1D Cervarix®) | 18-21 Year Old Women (3D Gardasil-4®) | 22-25 Year Old Women (3D Gardasil-4®)
Number analyzed (Participants) | 211 | 336 | 229 | 142
Participants | 211 | 335 | 229 | 142
Statistical Analysis 1: Comparison: 12-14-year-old Girls (1D Cervarix®) vs 22-25 Year Old Women (3D Gardasil-4®); NOTE: Younger one-dose recipients (9-11 Year Old Girls) and three-dose recipients (18-21 Year Old Women) both had a 100% seroconversion proportion for HPV16 at 24months, so a p-value for the difference of the seroconversion rate between them could not be calculated. Therefore, we only include the calculated p-value for the comparison of the seroconversion rate between older one-dose recipients (9-11 Year Old Girls) and three-dose recipients (22-25 Year Old Women); Test type: Equivalence — We will use a Fisher Exact test to test for the difference of the seroconversion rate between the older one-dose recipients and the older three-dose recipients; p = 1.000, Fisher Exact — A p-value under 0.05 will be regarded as significant

50. Secondary Outcome: Number Seropositive for HPV18 at 24 Months, By Enrollment Age Group
Description: as for outcome 7
Time Frame: 24 months
Population: The primary cohort for the analysis of HPV18 at 24 months by enrollment age group includes participants who received the appropriate number of vaccine doses within the specified windows, were initially seronegative for HPV18, underwent blood collection at the 24-month mark, and reported no additional HPV vaccinations outside the study before the 24-month blood collection, as confirmed by self-report or serologic testing for HPV6/HPV11.
Measure: Count of Participants; unit: Participants
Arm/Group | 9-11 Year Old Girls (1D Cervarix®) | 12-14-year-old Girls (1D Cervarix®) | 18-21 Year Old Women (3D Gardasil-4®) | 22-25 Year Old Women (3D Gardasil-4®)
Number analyzed (Participants) | 206 | 324 | 213 | 163
Participants | 205 | 316 | 208 | 159

51. Secondary Outcome: Comparison of GMCs for HPV18 Antibodies, Assessed at 24 Months, by Enrollment Age Group
Description: To evaluate whether age is associated with GMCs for HPV18 antibodies, assessed at 24 months after initial vaccination.
Time Frame: 24 month
Population: The cohort for the analysis of HPV18 at 24 months by enrollment age group includes participants who received the appropriate number of vaccine doses within the specified windows, were initially seronegative for HPV18, underwent blood collection at the 24-month mark, and reported no additional HPV vaccinations outside the study before the 24-month blood collection, as confirmed by self-report or serologic testing for HPV6/HPV11.
Measure: Geometric Mean (95% Confidence Interval); unit: International units (IU/mL)
Arm/Group | 9-11 Year Old Girls (1D Cervarix®) | 12-14-year-old Girls (1D Cervarix®) | 18-21 Year Old Women (3D Gardasil-4®) | 22-25 Year Old Women (3D Gardasil-4®)
Number analyzed (Participants) | 205 | 316 | 208 | 159
International units (IU/mL) | 8.4 [7.4 to 9.5] | 7.6 [6.8 to 8.5] | 9.9 [8.5 to 11.5] | 7.6 [6.5 to 8.9]
Statistical Analysis 1: Comparison: 9-11 Year Old Girls (1D Cervarix®) vs 18-21 Year Old Women (3D Gardasil-4®); [analysis description as in outcome 42, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 24, analysis 1]; GMC Ratio = 0.85, 99% CI 2-sided [0.65 to 1.10]
Statistical Analysis 2: Comparison: 12-14-year-old Girls (1D Cervarix®) vs 22-25 Year Old Women (3D Gardasil-4®); [analysis description as in outcome 42, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 24, analysis 1]; GMC Ratio = 1.00, 99% CI 2-sided [0.77 to 1.29]
Statistical Analysis 3: Comparison: 9-11 Year Old Girls (1D Cervarix®) vs 12-14-year-old Girls (1D Cervarix®) vs 18-21 Year Old Women (3D Gardasil-4®) vs 22-25 Year Old Women (3D Gardasil-4®); Test type: Equivalence — The p-values test for heterogeneity in the GMC ratios estimated from the stratified analyses; p = 0.24, The p-values test for heterogeneity — A p-value <0.05 is interpreted as significantly different GMC ratios in different strata

52. Secondary Outcome: Comparison of Seroconversion Proportions for HPV18, Assessed at 24 Months, by Enrollment Age Group
Description: as for outcome 49
Time Frame: 24 month
Population: as for outcome 51
Measure: Count of Participants; unit: Participants
Arm/Group | 9-11 Year Old Girls (1D Cervarix®) | 12-14-year-old Girls (1D Cervarix®) | 18-21 Year Old Women (3D Gardasil-4®) | 22-25 Year Old Women (3D Gardasil-4®)
Number analyzed (Participants) | 206 | 324 | 213 | 163
Participants | 205 | 316 | 208 | 159
Statistical Analysis 1: Comparison: 9-11 Year Old Girls (1D Cervarix®) vs 18-21 Year Old Women (3D Gardasil-4®); The calculated p-value for the comparison of the seroconversion rate of HPV18 at 24 months between younger one-dose recipients (9-12 Year Old Girls) and younger three-dose recipients (18-21 Year Old Women); Test type: Equivalence — We will use a Fisher Exact test to test for the difference of the seroconversion rate between younger one-dose and younger three-dose recipients; p = 0.216, Fisher Exact — A p-value under 0.05 will be regarded as significant
Statistical Analysis 2: Comparison: 12-14-year-old Girls (1D Cervarix®) vs 22-25 Year Old Women (3D Gardasil-4®); The calculated p-value for the comparison of the seroconversion rate of HPV18 at 24 months between older one-dose recipients (12-14 Year Old Girls) and older three-dose recipients (22-25 Year Old Women); Test type: Equivalence — We will use a Fisher Exact test to test for the difference of the seroconversion rate between older one-dose and older three-dose recipients; p = 1.000, Fisher Exact — A p-value under 0.05 will be regarded as significant

53. Secondary Outcome: Number Seropositive for HPV16, Assessed at 36 Months, by Enrollment Month Group
Description: HPV16 ELISA results at 36-months (final analysis) by arm in according to protocol (ATP) analytical cohort, stratified by enrollment month
Time Frame: 36 month
Population: The cohort for the analysis of HPV16 at 36 months by enrollment month grouping includes participants who received the appropriate number of vaccine doses within the specified windows, were initially seronegative for HPV16, underwent blood collection at the 36-month mark, and reported no additional HPV vaccinations outside the study before the 36-month blood collection, as confirmed by self-report or serologic testing for HPV6/HPV11.
Measure: Count of Participants; unit: Participants
Groups:
- Girls (1D Cervarix) Enrolled April-May; Girls (1D Cervarix) Enrolled June-August: Participants 9-14 years old receive Cervarix IM at baseline. Recombinant Human Papillomavirus Bivalent Vaccine: Given IM
- Women (3D Gardasil) Enrolled April-May; Women (3D Gardasil) Enrolled June-August: Participants 18-25 years old receive Gardasil IM at baseline and at 2 and 6 months in the absence of unacceptable toxicity. Quadrivalent Human Papillomavirus (types 6, 11, 16, 18) Recombinant Vaccine: Given IM
Arm/Group | Girls (1D Cervarix) Enrolled April-May | Women (3D Gardasil) Enrolled April-May | Girls (1D Cervarix) Enrolled June-August | Women (3D Gardasil) Enrolled June-August
Number analyzed (Participants) | 195 | 145 | 344 | 221
Participants | 195 | 145 | 343 | 221

54. Secondary Outcome: Comparison of GMCs for HPV16 Antibodies Assessed at 36 Months, by Enrollment Month Group
Description: as for outcome 53
Time Frame: 36 month
Population: as for outcome 53
Measure: Geometric Mean (95% Confidence Interval); unit: International units (IU/mL)
Arm/Group | Girls (1D Cervarix) Enrolled April-May | Women (3D Gardasil) Enrolled April-May | Girls (1D Cervarix) Enrolled June-August | Women (3D Gardasil) Enrolled June-August
Number analyzed (Participants) | 195 | 145 | 343 | 221
International units (IU/mL) | 21.6 [18.8 to 24.8] | 41.6 [36.3 to 47.7] | 21.3 [19.2 to 23.6] | 43.6 [38.2 to 49.7]
Statistical Analysis 1: Comparison: Girls (1D Cervarix) Enrolled April-May vs Women (3D Gardasil) Enrolled April-May; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 18, analysis 1]; GMC Ratio = 0.52, 96% CI 2-sided [0.43 to 0.64]
Statistical Analysis 2: Comparison: Girls (1D Cervarix) Enrolled June-August vs Women (3D Gardasil) Enrolled June-August; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 18, analysis 1]; GMC Ratio = 0.49, 96% CI 2-sided [0.41 to 0.58]
Statistical Analysis 3: Comparison: Girls (1D Cervarix) Enrolled April-May vs Women (3D Gardasil) Enrolled April-May vs Girls (1D Cervarix) Enrolled June-August vs Women (3D Gardasil) Enrolled June-August; Test type: Equivalence — The p-values test for heterogeneity in the GMC ratios estimated from the stratified analyses; p = 0.73, The p-values test for heterogeneity — A p-value <0.05 is interpreted as significantly different GMC ratios in different strata

55. Secondary Outcome: Comparison of Seroconversion Proportions for HPV16, Assessed at 36 Months, by Enrollment Month
Description: as for outcome 53
Time Frame: 36 month
Population: The primary cohort for the analysis of HPV16 at 36 months includes participants who received the appropriate number of vaccine doses within the specified windows, were initially seronegative for HPV16, underwent blood collection at the 36-month mark, and reported no additional HPV vaccinations outside the study before the 36-month blood collection, as confirmed by self-report or serologic testing for HPV6/HPV11.
Measure: Count of Participants; unit: Participants
Arm/Group | Girls (1D Cervarix) Enrolled April-May | Women (3D Gardasil) Enrolled April-May | Girls (1D Cervarix) Enrolled June-August | Women (3D Gardasil) Enrolled June-August
Number analyzed (Participants) | 195 | 145 | 344 | 221
Participants | 195 | 145 | 343 | 221
Statistical Analysis 1: Comparison: Girls (1D Cervarix) Enrolled June-August vs Women (3D Gardasil) Enrolled June-August; NOTE: One-dose recipients and three-dose recipients enrolled April - May both had a 100% seroconversion proportion for HPV16 at 36 months, so the p-value for the difference of the seroconversion rate between them could not be calculated. Therefore, we only include the calculated p-value for the comparison of the seroconversion rate between one-dose recipients and three-dose recipients enrolled June - August; Test type: Equivalence — We will use a Fisher Exact test to test for the difference of the seroconversion rate one-dose and three-dose recipients who enrolled June - August; p = 1.000, Fisher Exact — A p-value under 0.05 will be regarded as significant

56. Secondary Outcome: Number Seropositive for HPV18, Assessed at 36 Months, by Enrollment Month Group
Description: HPV18 ELISA results at 36-months (final analysis) by arm in according to protocol (ATP) analytical cohort, stratified by enrollment month
Time Frame: 36 month
Population: The cohort for the analysis of HPV18 at 36 months by enrollment month grouping includes participants who received the appropriate number of vaccine doses within the specified windows, were initially seronegative for HPV18, underwent blood collection at the 36-month mark, and reported no additional HPV vaccinations outside the study before the 36-month blood collection, as confirmed by self-report or serologic testing for HPV6/HPV11.
Measure: Count of Participants; unit: Participants
Arm/Group | Girls (1D Cervarix) Enrolled April-May | Women (3D Gardasil) Enrolled April-May | Girls (1D Cervarix) Enrolled June-August | Women (3D Gardasil) Enrolled June-August
Number analyzed (Participants) | 184 | 154 | 339 | 219
Participants | 182 | 149 | 335 | 209

57. Secondary Outcome: Comparison of GMCs for HPV18 Antibodies, Assessed at 36 Months, by Enrollment Month Group
Description: as for outcome 56
Time Frame: 36 month
Population: as for outcome 56
Measure: Geometric Mean (95% Confidence Interval); unit: International units (IU/mL)
Arm/Group | Girls (1D Cervarix) Enrolled April-May | Women (3D Gardasil) Enrolled April-May | Girls (1D Cervarix) Enrolled June-August | Women (3D Gardasil) Enrolled June-August
Number analyzed (Participants) | 182 | 149 | 335 | 209
International units (IU/mL) | 7.9 [6.8 to 9.1] | 6.3 [5.3 to 7.4] | 8.1 [7.3 to 9.1] | 8.0 [6.8 to 9.4]
Statistical Analysis 1: Comparison: Girls (1D Cervarix) Enrolled April-May vs Women (3D Gardasil) Enrolled April-May; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 18, analysis 1]; GMC Ratio = 1.26, 96% CI [1.00 to 1.58]
Statistical Analysis 2: Comparison: Girls (1D Cervarix) Enrolled June-August vs Women (3D Gardasil) Enrolled June-August; Test type: Non-Inferiority — [test comment as in outcome 18, analysis 1]; GMC Ratio = 1.01, 96% CI [0.83 to 1.24]
Statistical Analysis 3: Comparison: Girls (1D Cervarix) Enrolled April-May vs Women (3D Gardasil) Enrolled April-May vs Girls (1D Cervarix) Enrolled June-August vs Women (3D Gardasil) Enrolled June-August; Test type: Equivalence — The p-values test for heterogeneity in the GMC ratios estimated from the stratified analyses; p = 0.15, The p-values test for heterogeneity — A p-value <0.05 is interpreted as significantly different GMC ratios in different strata

58. Secondary Outcome: Comparison of Seroconversion Proportions for HPV18, Assessed at 36 Months, by Enrollment Month
Description: as for outcome 56
Time Frame: 36 month
Population: as for outcome 56
Measure: Count of Participants; unit: Participants
Arm/Group | Girls (1D Cervarix) Enrolled April-May | Women (3D Gardasil) Enrolled April-May | Girls (1D Cervarix) Enrolled June-August | Women (3D Gardasil) Enrolled June-August
Number analyzed (Participants) | 184 | 154 | 339 | 219
Participants | 182 | 149 | 335 | 209
Statistical Analysis 1: Comparison: Girls (1D Cervarix) Enrolled April-May vs Women (3D Gardasil) Enrolled April-May; The calculated p-value for the comparison of the seroconversion rate of HPV18 at 36 months between one-dose recipients and three-dose recipients enrolled April - May; Test type: Equivalence — We will use a Fisher Exact test to test for the difference of the seroconversion rate between one-dose and three-dose recipients enrolled April - May; p = 0.253, Fisher Exact — A p-value under 0.05 will be regarded as significant
Statistical Analysis 2: Comparison: Girls (1D Cervarix) Enrolled June-August vs Women (3D Gardasil) Enrolled June-August; The calculated p-value for the comparison of the seroconversion rate of HPV18 at 36 months between one-dose recipients and three-dose recipients enrolled June - August; Test type: Equivalence — We will use a Fisher Exact test to test for the difference of the seroconversion rate between one-dose and three-dose recipients enrolled June - August; p = 0.015, Fisher Exact — A p-value under 0.05 will be regarded as significant

59. Secondary Outcome: Number Seropositive for HPV16, Assessed at 24 Months, by Enrollment Month
Description: HPV16 ELISA results at 24-months (interim analysis) by arm in according to protocol (ATP) analytical cohort, stratified by enrollment month
Time Frame: 24 month
Population: The cohort for the analysis of HPV16 at 24 months by enrollment month grouping includes participants who received the appropriate number of vaccine doses within the specified windows, were initially seronegative for HPV16, underwent blood collection at the 24-month mark, and reported no additional HPV vaccinations outside the study before the 36-month blood collection, as confirmed by self-report or serologic testing for HPV6/HPV11.
Measure: Count of Participants; unit: Participants
Arm/Group | Girls (1D Cervarix) Enrolled April-May | Women (3D Gardasil) Enrolled April-May | Girls (1D Cervarix) Enrolled June-August | Women (3D Gardasil) Enrolled June-August
Number analyzed (Participants) | 196 | 147 | 351 | 224
Participants | 196 | 147 | 350 | 224

60. Secondary Outcome: Comparison of GMCs for HPV16 Antibodies Assessed at 24 Months, by Enrollment Month Group
Description: as for outcome 59
Time Frame: 24 month
Population: The cohort for the analysis of HPV16 at 24 months by enrollment month grouping includes participants who received the appropriate number of vaccine doses within the specified windows, were initially seronegative for HPV16, underwent blood collection at the 24-month mark, and reported no additional HPV vaccinations outside the study before the 24-month blood collection, as confirmed by self-report or serologic testing for HPV6/HPV11.
Measure: Geometric Mean (95% Confidence Interval); unit: International units (IU/mL)
Arm/Group | Girls (1D Cervarix) Enrolled April-May | Women (3D Gardasil) Enrolled April-May | Girls (1D Cervarix) Enrolled June-August | Women (3D Gardasil) Enrolled June-August
Number analyzed (Participants) | 196 | 147 | 350 | 224
International units (IU/mL) | 20.4 [17.9 to 23.4] | 47.9 [41.8 to 54.8] | 20.7 [18.7 to 22.9] | 49.2 [43.4 to 55.9]
Statistical Analysis 1: Comparison: Girls (1D Cervarix) Enrolled April-May vs Women (3D Gardasil) Enrolled April-May; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 24, analysis 1]; GMC Ratio = 0.43, 99% CI [0.33 to 0.55]
Statistical Analysis 2: Comparison: Girls (1D Cervarix) Enrolled June-August vs Women (3D Gardasil) Enrolled June-August; Test type: Non-Inferiority — [test comment as in outcome 24, analysis 1]; GMC Ratio = 0.42, 99% CI 2-sided [0.34 to 0.52]
Statistical Analysis 3: Comparison: Girls (1D Cervarix) Enrolled April-May vs Women (3D Gardasil) Enrolled April-May vs Girls (1D Cervarix) Enrolled June-August vs Women (3D Gardasil) Enrolled June-August; Test type: Equivalence — The p-values test for heterogeneity in the GMC ratios estimated from the stratified analyses; p = 0.95, p-values test for heterogeneity — A p-value <0.05 is interpreted as significantly different GMC ratios in different strata

61. Secondary Outcome: Comparison of Seroconversion Proportions for HPV16, Assessed at 24 Months, by Enrollment Month
Description: as for outcome 59
Time Frame: 24 month
Population: as for outcome 60
Measure: Count of Participants; unit: Participants
Arm/Group | Girls (1D Cervarix) Enrolled April-May | Women (3D Gardasil) Enrolled April-May | Girls (1D Cervarix) Enrolled June-August | Women (3D Gardasil) Enrolled June-August
Number analyzed (Participants) | 196 | 147 | 351 | 224
Participants | 196 | 147 | 350 | 224
Statistical Analysis 1: Comparison: Girls (1D Cervarix) Enrolled June-August vs Women (3D Gardasil) Enrolled June-August; NOTE: One-dose recipients and three-dose recipients enrolled April - May both had a 100% seroconversion proportion for HPV16 at 24 months, so the p-value for the difference of the seroconversion rate between them could not be calculated. Therefore, we only include the calculated p-value for the comparison of the seroconversion rate between one-dose recipients and three-dose recipients enrolled June - August; Test type: Equivalence — [test comment as in outcome 58, analysis 2]; p = 1.000, Fisher Exact — A p-value under 0.05 will be regarded as significant

62. Secondary Outcome: Number Seropositive for HPV18, Assessed at 24 Months, by Enrollment Month Group
Description: HPV18 ELISA results at 24-months (interim analysis) by arm in according to protocol (ATP) analytical cohort, stratified by enrollment month
Time Frame: 24 month
Population: The cohort for the analysis of HPV18 at 24 months by enrollment month grouping includes participants who received the appropriate number of vaccine doses within the specified windows, were initially seronegative for HPV18, underwent blood collection at the 24-month mark, and reported no additional HPV vaccinations outside the study before the 24-month blood collection, as confirmed by self-report or serologic testing for HPV6/HPV11.
Measure: Count of Participants; unit: Participants
Arm/Group | Girls (1D Cervarix) Enrolled April-May | Women (3D Gardasil) Enrolled April-May | Girls (1D Cervarix) Enrolled June-August | Women (3D Gardasil) Enrolled June-August
Number analyzed (Participants) | 185 | 155 | 345 | 221
Participants | 182 | 154 | 339 | 213

63. Secondary Outcome: Comparison of GMCs for HPV18 Antibodies Assessed at 24 Months, by Enrollment Month Group
Description: as for outcome 62
Time Frame: 24 month
Population: as for outcome 62
Measure: Geometric Mean (95% Confidence Interval); unit: International units (IU/mL)
Arm/Group | Girls (1D Cervarix) Enrolled April-May | Women (3D Gardasil) Enrolled April-May | Girls (1D Cervarix) Enrolled June-August | Women (3D Gardasil) Enrolled June-August
Number analyzed (Participants) | 182 | 154 | 339 | 213
International units (IU/mL) | 7.4 [6.5 to 8.5] | 8.2 [7.0 to 9.6] | 8.2 [7.4 to 9.2] | 9.3 [7.9 to 10.8]
Statistical Analysis 1: Comparison: Girls (1D Cervarix) Enrolled April-May vs Women (3D Gardasil) Enrolled April-May; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 24, analysis 1]; GMC Ratio = 0.91, 99% CI 2-sided [0.69 to 1.19]
Statistical Analysis 2: Comparison: Girls (1D Cervarix) Enrolled June-August vs Women (3D Gardasil) Enrolled June-August; Test type: Non-Inferiority — [test comment as in outcome 24, analysis 1]; GMC Ratio = 0.89, 99% CI 2-sided [0.69 to 1.14]
Statistical Analysis 3: Comparison: Girls (1D Cervarix) Enrolled April-May vs Women (3D Gardasil) Enrolled April-May vs Girls (1D Cervarix) Enrolled June-August vs Women (3D Gardasil) Enrolled June-August; Test type: Equivalence — The p-values test for heterogeneity in the GMC ratios estimated from the stratified analyses; p = 0.88, p-values test for heterogeneity — A p-value <0.05 is interpreted as significantly different GMC ratios in different strata

64. Secondary Outcome: Comparison of Seroconversion Proportions for HPV18, Assessed at 24 Months, by Enrollment Month
Description: as for outcome 62
Time Frame: 24 month
Population: as for outcome 62
Measure: Count of Participants; unit: Participants
Arm/Group | Girls (1D Cervarix) Enrolled April-May | Women (3D Gardasil) Enrolled April-May | Girls (1D Cervarix) Enrolled June-August | Women (3D Gardasil) Enrolled June-August
Number analyzed (Participants) | 185 | 155 | 345 | 221
Participants | 182 | 154 | 339 | 213
Statistical Analysis 1: Comparison: Girls (1D Cervarix) Enrolled April-May vs Women (3D Gardasil) Enrolled April-May; The calculated p-value for the comparison of the seroconversion rate of HPV18 at 24 months between one-dose recipients and three-dose recipients enrolled April - May; Test type: Equivalence — [test comment as in outcome 58, analysis 1]; p = 0.629, Fisher Exact — A p-value under 0.05 will be regarded as significant
Statistical Analysis 2: Comparison: Girls (1D Cervarix) Enrolled June-August vs Women (3D Gardasil) Enrolled June-August; The calculated p-value for the comparison of the seroconversion rate of HPV18 at 24 months between one-dose recipients and three-dose recipients enrolled June - August; Test type: Equivalence — [test comment as in outcome 58, analysis 2]; p = 0.175, Fisher Exact — A p-value under 0.05 will be regarded as significant

65. Secondary Outcome: Number Seropositive for HPV16, Assessed at 36 Months, by Enrollment District
Description: HPV16 ELISA results at 36-months (final analysis) by arm in the according to protocol analytical cohort stratified by enrollment region.
Time Frame: 36 month
Population: The cohort for the analysis of HPV16 at 36 months by enrollment district grouping includes participants who received the appropriate number of vaccine doses within the specified windows, were initially seronegative for HPV16, underwent blood collection at the 36-month mark, and reported no additional HPV vaccinations outside the study before the 36-month blood collection, as confirmed by self-report or serologic testing for HPV6/HPV11.
Measure: Count of Participants; unit: Participants
Groups:
- Coastal Girls (1D Cervarix); Mountainous Girls (1D Cervarix): Participants 9-14 years old receive Cervarix IM at baseline. Recombinant Human Papillomavirus Bivalent Vaccine: Given IM
- Coastal Women (3D Gardasil); Mountainous Women (3D Gardasil): Participants 18-25 years old receive Gardasil IM at baseline and at 2 and 6 months in the absence of unacceptable toxicity. Quadrivalent Human Papillomavirus (types 6, 11, 16, 18) Recombinant Vaccine: Given IM
Arm/Group | Coastal Girls (1D Cervarix) | Coastal Women (3D Gardasil) | Mountainous Girls (1D Cervarix) | Mountainous Women (3D Gardasil)
Number analyzed (Participants) | 250 | 169 | 289 | 197
Participants | 249 | 169 | 289 | 197

66. Secondary Outcome: Comparison of GMCs for HPV16 Antibodies, Assessed at 36 Months, by Enrollment District
Description: as for outcome 65
Time Frame: 36 month
Population: The cohort for the analysis of HPV16 at 36 months by district grouping includes participants who received the appropriate number of vaccine doses within the specified windows, were initially seronegative for HPV16, underwent blood collection at the 36-month mark, and reported no additional HPV vaccinations outside the study before the 36-month blood collection, as confirmed by self-report or serologic testing for HPV6/HPV11.
Measure: Geometric Mean (95% Confidence Interval); unit: International units (IU/mL)
Arm/Group | Coastal Girls (1D Cervarix) | Coastal Women (3D Gardasil) | Mountainous Girls (1D Cervarix) | Mountainous Women (3D Gardasil)
Number analyzed (Participants) | 249 | 169 | 289 | 197
International units (IU/mL) | 21.5 [19.0 to 24.3] | 41.0 [35.7 to 47.1] | 21.4 [19.1 to 24.0] | 44.6 [38.9 to 51.0]
Statistical Analysis 1: Comparison: Coastal Girls (1D Cervarix) vs Coastal Women (3D Gardasil); [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 18, analysis 1]; GMC Ratio = 0.52, 96% CI [0.43 to 0.64]
Statistical Analysis 2: Comparison: Mountainous Girls (1D Cervarix) vs Mountainous Women (3D Gardasil); Test type: Non-Inferiority — [test comment as in outcome 18, analysis 1]; GMC Ratio = 0.48, 96% CI [0.40 to 0.58]
Statistical Analysis 3: Comparison: Coastal Girls (1D Cervarix) vs Coastal Women (3D Gardasil) vs Mountainous Girls (1D Cervarix) vs Mountainous Women (3D Gardasil); Test type: Equivalence — The p-values test for heterogeneity in the GMC ratios estimated from the stratified analyses; p = 0.46, p-values test for heterogeneity — A p-value <0.05 is interpreted as significantly different GMC ratios in different strata

67. Secondary Outcome: Comparison of Seroconversion Proportions for HPV16, Assessed at 36 Months, by Enrollment District
Description: as for outcome 65
Time Frame: 36 month
Population: as for outcome 66
Measure: Median (95% Confidence Interval); unit: International units (IU/mL)
Arm/Group | Coastal Girls (1D Cervarix) | Coastal Women (3D Gardasil) | Mountainous Girls (1D Cervarix) | Mountainous Women (3D Gardasil)
Number analyzed (Participants) | 250 | 169 | 289 | 197
International units (IU/mL) | 99.6 [98.1 to 100.0] | 100.0 [98.2 to 100.0] | 100.0 [99.0 to 100.0] | 100.0 [98.5 to 100.0]
Statistical Analysis 1: Comparison: Coastal Girls (1D Cervarix) vs Coastal Women (3D Gardasil); NOTE: One-dose recipients and three-dose recipients enrolled from mountainous districts both had a 100% seroconversion proportion for HPV16 at 36 months, so the p-value for the difference of the seroconversion rate between them could not be calculated. Therefore, we only include the calculated p-value for the comparison of the seroconversion rate for HPV16 at 36 months between one-dose recipients and three-dose recipients enrolled from coastal districts; Test type: Equivalence — We will use a Fisher Exact test to test for the difference of the seroconversion rate between one-dose and three-dose recipients from coastal districts; p = 1.000, Fisher Exact — A p-value under 0.05 will be regarded as significant

68. Secondary Outcome: Number Seropositive for HPV18, Assessed at 36 Months, by Enrollment District
Description: HPV18 ELISA results at 36-months (final analysis) by arm in the according to protocol analytical cohort stratified by enrollment region.
Time Frame: 36 month
Population: The cohort for the analysis of HPV18 at 36 months by district grouping includes participants who received the appropriate number of vaccine doses within the specified windows, were initially seronegative for HPV18, underwent blood collection at the 36-month mark, and reported no additional HPV vaccinations outside the study before the 36-month blood collection, as confirmed by self-report or serologic testing for HPV6/HPV11.
Measure: Count of Participants; unit: Participants
Arm/Group | Coastal Girls (1D Cervarix) | Coastal Women (3D Gardasil) | Mountainous Girls (1D Cervarix) | Mountainous Women (3D Gardasil)
Number analyzed (Participants) | 244 | 163 | 279 | 210
Participants | 240 | 157 | 277 | 201

69. Secondary Outcome: Comparison of GMCs for HPV18 Antibodies, Assessed at 36 Months, by Enrollment District
Description: as for outcome 68
Time Frame: 36 month
Population: as for outcome 68
Measure: Geometric Mean (95% Confidence Interval); unit: International units (IU/mL)
Arm/Group | Coastal Girls (1D Cervarix) | Coastal Women (3D Gardasil) | Mountainous Girls (1D Cervarix) | Mountainous Women (3D Gardasil)
Number analyzed (Participants) | 240 | 157 | 277 | 201
International units (IU/mL) | 8.5 [7.5 to 9.5] | 6.7 [5.7 to 7.8] | 7.7 [6.8 to 8.7] | 7.7 [6.6 to 9.1]
Statistical Analysis 1: Comparison: Coastal Girls (1D Cervarix) vs Coastal Women (3D Gardasil); [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 18, analysis 1]; GMC Ratio = 1.27, 96% CI [1.03 to 1.57]
Statistical Analysis 2: Comparison: Mountainous Girls (1D Cervarix) vs Mountainous Women (3D Gardasil); Test type: Non-Inferiority — [test comment as in outcome 18, analysis 1]; GMC Ratio = 0.99, 96% CI [0.80 to 1.23]
Statistical Analysis 3: Comparison: Coastal Girls (1D Cervarix) vs Coastal Women (3D Gardasil) vs Mountainous Girls (1D Cervarix) vs Mountainous Women (3D Gardasil); Test type: Equivalence — The p-values test for heterogeneity in the GMC ratios estimated from the stratified analyses; p = 0.095, p-values test for heterogeneity — A p-value <0.05 is interpreted as significantly different GMC ratios in different strata

70. Secondary Outcome: Comparison of Seroconversion Proportions for HPV18, Assessed at 36 Months, by Enrollment District
Description: as for outcome 68
Time Frame: 36 month
Population: The cohort for the analysis of HPV18 at 36 months by enrollment district grouping includes participants who received the appropriate number of vaccine doses within the specified windows, were initially seronegative for HPV18, underwent blood collection at the 36-month mark, and reported no additional HPV vaccinations outside the study before the 36-month blood collection, as confirmed by self-report or serologic testing for HPV6/HPV11.
Measure: Count of Participants; unit: Participants
Arm/Group | Coastal Girls (1D Cervarix) | Coastal Women (3D Gardasil) | Mountainous Girls (1D Cervarix) | Mountainous Women (3D Gardasil)
Number analyzed (Participants) | 244 | 163 | 279 | 210
Participants | 240 | 157 | 277 | 201
Statistical Analysis 1: Comparison: Coastal Girls (1D Cervarix) vs Coastal Women (3D Gardasil); The calculated p-value for the comparison of the seroconversion rate for HPV18 at 36 months between one-dose recipients and three-dose recipients enrolled from coastal districts; Test type: Equivalence — We will use a Fisher Exact test to test for the difference of the seroconversion rate between one-dose and three-dose recipients enrolled from coastal districts; p = 0.327, Fisher Exact — A p-value under 0.05 will be regarded as significant
Statistical Analysis 2: Comparison: Mountainous Girls (1D Cervarix) vs Mountainous Women (3D Gardasil); The calculated p-value for the comparison of the seroconversion rate for HPV18 at 36 months between one-dose recipients and three-dose recipients enrolled from mountainous districts; Test type: Equivalence — We will use a Fisher Exact test to test for the difference of the seroconversion rate between one-dose and three-dose recipients enrolled from mountainous districts; p = 0.012, Fisher Exact — A p-value under 0.05 will be regarded as significant

71. Secondary Outcome: Number Seropositive for HPV16, Assessed at 24 Months, by Enrollment District
Description: HPV16 ELISA results at 24-months (interim analysis) by arm in the according to protocol analytical cohort stratified by enrollment region.
Time Frame: 24 month
Population: The cohort for the analysis of HPV16 at 24 months by district grouping includes participants who received the appropriate number of vaccine doses within the specified windows, were initially seronegative for HPV16, underwent blood collection at the 24-month mark, and reported no additional HPV vaccinations outside the study before the 24-month blood collection, as confirmed by self-report or serologic testing for HPV6/HPV11.
Measure: Count of Participants; unit: Participants
Arm/Group | Coastal Girls (1D Cervarix) | Coastal Women (3D Gardasil) | Mountainous Girls (1D Cervarix) | Mountainous Women (3D Gardasil)
Number analyzed (Participants) | 254 | 171 | 293 | 200
Participants | 253 | 171 | 293 | 200

72. Secondary Outcome: Comparison of GMCs for HPV16 Antibodies, Assessed at 24 Months, by Enrollment District
Description: as for outcome 71
Time Frame: 24 month
Population: as for outcome 71
Measure: Geometric Mean (95% Confidence Interval); unit: International units (IU/mL)
Arm/Group | Coastal Girls (1D Cervarix) | Coastal Women (3D Gardasil) | Mountainous Girls (1D Cervarix) | Mountainous Women (3D Gardasil)
Number analyzed (Participants) | 253 | 171 | 293 | 200
International units (IU/mL) | 21.0 [18.5 to 23.7] | 46.3 [40.5 to 53.0] | 20.3 [18.3 to 22.7] | 51.1 [44.8 to 58.4]
Statistical Analysis 1: Comparison: Coastal Girls (1D Cervarix) vs Coastal Women (3D Gardasil); Test type: Non-Inferiority — [test comment as in outcome 24, analysis 1]; GMC Ratio = 0.45, 99% CI 2-sided [0.36 to 0.58]
Statistical Analysis 2: Comparison: Mountainous Girls (1D Cervarix) vs Mountainous Women (3D Gardasil); Test type: Non-Inferiority — [test comment as in outcome 24, analysis 1]; GMC Ratio = 0.40, 99% CI 2-sided [0.32 to 0.50]
Statistical Analysis 3: Comparison: Coastal Girls (1D Cervarix) vs Coastal Women (3D Gardasil) vs Mountainous Girls (1D Cervarix) vs Mountainous Women (3D Gardasil); Test type: Equivalence — The p-values test for heterogeneity in the GMC ratios estimated from the stratified analyses; p = 0.30, p-values test for heterogeneity — A p-value <0.05 is interpreted as significantly different GMC ratios in different strata

73. Secondary Outcome: Comparison of Seroconversion Proportions for HPV16, Assessed at 24 Months, by Enrollment District
Description: as for outcome 71
Time Frame: 24 month
Population: as for outcome 71
Measure: Count of Participants; unit: Participants
Arm/Group | Coastal Girls (1D Cervarix) | Coastal Women (3D Gardasil) | Mountainous Girls (1D Cervarix) | Mountainous Women (3D Gardasil)
Number analyzed (Participants) | 254 | 171 | 293 | 200
Participants | 253 | 171 | 293 | 200
Statistical Analysis 1: Comparison: Coastal Girls (1D Cervarix) vs Coastal Women (3D Gardasil); NOTE: One-dose recipients and three-dose recipients enrolled from mountainous districts had a 100% seroconversion proportion for HPV16 at 24 months, so the p-value for the difference of the seroconversion rate between them could not be calculated. Therefore, we only include the calculated p-value for the comparison of the seroconversion rate for HPV16 at 24 months between one-dose recipients and three-dose recipients enrolled from coastal districts; Test type: Equivalence — [test comment as in outcome 70, analysis 1]; p = 1.000, Fisher Exact — A p-value under 0.05 will be regarded as significant

74. Secondary Outcome: Number Seropositive for HPV18, Assessed at 24 Months, by Enrollment District
Description: HPV18 ELISA results at 24-months (interim analysis) by arm in the according to protocol analytical cohort stratified by enrollment region.
Time Frame: 24 month
Population: The cohort for the analysis of HPV18 at 24 months by district grouping includes participants who received the appropriate number of vaccine doses within the specified windows, were initially seronegative for HPV18, underwent blood collection at the 24-month mark, and reported no additional HPV vaccinations outside the study before the 24-month blood collection, as confirmed by self-report or serologic testing for HPV6/HPV11.
Measure: Count of Participants; unit: Participants
Arm/Group | Coastal Girls (1D Cervarix) | Coastal Women (3D Gardasil) | Mountainous Girls (1D Cervarix) | Mountainous Women (3D Gardasil)
Number analyzed (Participants) | 247 | 164 | 283 | 212
Participants | 242 | 161 | 279 | 206

75. Secondary Outcome: Comparison of GMCs for HPV18 Antibodies, Assessed at 24 Months, by Enrollment District
Description: as for outcome 74
Time Frame: 24 month
Population: as for outcome 74
Measure: Geometric Mean (95% Confidence Interval); unit: International units (IU/mL)
Arm/Group | Coastal Girls (1D Cervarix) | Coastal Women (3D Gardasil) | Mountainous Girls (1D Cervarix) | Mountainous Women (3D Gardasil)
Number analyzed (Participants) | 242 | 161 | 279 | 206
International units (IU/mL) | 8.4 [7.4 to 9.5] | 8.2 [7.0 to 9.5] | 7.6 [6.7 to 8.5] | 9.4 [8.0 to 11.0]
Statistical Analysis 1: Comparison: Coastal Girls (1D Cervarix) vs Coastal Women (3D Gardasil); [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 24, analysis 1]; GMC Ratio = 1.02, 99% CI [0.79 to 1.32]
Statistical Analysis 2: Comparison: Mountainous Girls (1D Cervarix) vs Mountainous Women (3D Gardasil); Test type: Non-Inferiority — [test comment as in outcome 24, analysis 1]; GMC Ratio = 0.81, 99% CI [0.63 to 1.04]
Statistical Analysis 3: Comparison: Coastal Girls (1D Cervarix) vs Coastal Women (3D Gardasil) vs Mountainous Girls (1D Cervarix) vs Mountainous Women (3D Gardasil); Test type: Equivalence — The p-values test for heterogeneity in the GMC ratios estimated from the stratified analyses; p = 0.10, p-values test for heterogeneity — A p-value <0.05 is interpreted as significantly different GMC ratios in different strata

76. Secondary Outcome: Comparison of Seroconversion Proportions for HPV18, Assessed at 24 Months, by Enrollment District
Description: as for outcome 74
Time Frame: 24 month
Population: as for outcome 74
Measure: Count of Participants; unit: Participants
Arm/Group | Coastal Girls (1D Cervarix) | Coastal Women (3D Gardasil) | Mountainous Girls (1D Cervarix) | Mountainous Women (3D Gardasil)
Number analyzed (Participants) | 247 | 164 | 283 | 212
Participants | 242 | 161 | 279 | 206
Statistical Analysis 1: Comparison: Coastal Girls (1D Cervarix) vs Coastal Women (3D Gardasil); The calculated p-value for the comparison of the seroconversion rate for HPV18 at 24 months between one-dose recipients and three-dose recipients enrolled from coastal districts; Test type: Equivalence — [test comment as in outcome 70, analysis 1]; p = 1.000, Fisher Exact — A p-value under 0.05 will be regarded as significant
Statistical Analysis 2: Comparison: Mountainous Girls (1D Cervarix) vs Mountainous Women (3D Gardasil); The calculated p-value for the comparison of the seroconversion rate for HPV18 at 24 months between one-dose recipients and three-dose recipients enrolled from mountainous districts; Test type: Equivalence — [test comment as in outcome 70, analysis 2]; p = 0.339, Fisher Exact — A p-value under 0.05 will be regarded as significant

ADVERSE EVENTS:
Time Frame: The time points and duration of assessment of adverse events differs for each participant according to their enrollment and exit dates. Systematic assessment of adverse events began the first vaccination date and ended 180 days after last vaccination date. Non-systematic assessment began 181 days after last vaccination and ends the date the participant exits the study. Some participants are not yet exited from the study; however, for these results, the end date is April 23, 2024.
Description: All adverse events, serious and not serious, were documented. Systematic assessment was done through inquiries at the study visit or contact following each vaccination. The clinician probed for adverse events by asking the participant whether she has been diagnosed with an illness, disabled for more than one day, or hospitalized since her last visit. Non-systematic assessment was done through spontaneous reports, including calls to a toll-free number.
Groups:
- Girls (1D Cervarix®) Systematic Collection Phase; Women (3D Gardasil-4®) Systematic Collection Phase: All adverse events, serious and not serious, were documented. Systematic assessment was done through inquiries at the study visit or contact following each vaccination. The clinician probed for adverse events by asking the participant whether she has been diagnosed with an illness, disabled for more than one day, or hospitalized since her last visit.
- Girls (1D Cervarix®) Non-systematic Collection Phase; Women (3D Gardasil-4®) Non-systematic Collection Phase: All adverse events, serious and not serious, were documented. Non-systematic assessment was done through spontaneous reports, including calls to a toll-free number.
Arm/Group | Girls (1D Cervarix®) Systematic Collection Phase | Women (3D Gardasil-4®) Systematic Collection Phase | Girls (1D Cervarix®) Non-systematic Collection Phase | Women (3D Gardasil-4®) Non-systematic Collection Phase
All-Cause Mortality (participants affected / at risk) | 0/620 | 1/620 | 1/620 | 0/620
Serious Adverse Events (participants affected / at risk) | 2/620 | 13/620 | 3/620 | 34/620
Other Adverse Events (participants affected / at risk) | 71/620 | 166/620 | 62/620 | 73/620
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Girls (1D Cervarix®) Systematic Collection Phase (N=620) | Women (3D Gardasil-4®) Systematic Collection Phase (N=620) | Girls (1D Cervarix®) Non-systematic Collection Phase (N=620) | Women (3D Gardasil-4®) Non-systematic Collection Phase (N=620)
Rhesus isoimmunization affecting management of mother (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Not related to vaccine
Ankyloglossia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Not related to vaccine
Acute appendicitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Not related to vaccine
Intrauterine contraceptive device complication (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Not related to vaccine
Alopecia areata (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Not related to vaccine
Asthma, unspecified (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Not related to vaccine
Acute endocarditis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Not related to vaccine
Meningitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Not related to vaccine
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Not related to vaccine
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Not related to vaccine
Urinary tract infection, site not specified (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Not related to vaccine
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Not related to vaccine
Uterine scar (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Not related to vaccine
Acute erythroid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Not related to vaccine
Malignant neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Not related to vaccine
Pituitary neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Not related to vaccine
Cerebrospinal fluid leakage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Not related to vaccine
Abortion spontaneous complete NOS (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 3 (3) | 0 (0) | 1 (1) — Not related to vaccine. NOTE: Event was collected by both systematic and non-systematic methods.
Abortion spontaneous incomplete (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Not related to vaccine
Blighted ovum (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 1 (1) — Not related to vaccine. NOTE: Event was collected by both systematic and non-systematic methods.
Breech presentation (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 3 (3) — Not related to vaccine
Diabetes in pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Not related to vaccine
Failed induction of labour (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 4 (4) — Not related to vaccine. NOTE: Event was collected by both systematic and non-systematic methods.
Failed trial of labour (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — Not related to vaccine
Foetopelvic disproportion (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Not related to vaccine
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 2 (2) — Not related to vaccine
Intra-uterine hypoxia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 2 (2) — Not related to vaccine
Large for dates baby (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 2 (2) — Not related to vaccine
Missed abortion (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Not related to vaccine
Obstructed labour, unspecified (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Not related to vaccine
Oligohydramnios (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Not related to vaccine
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Not related to vaccine
Threatened abortion (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Not related to vaccine
Transverse presentation (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 2 (2) — Not related to vaccine
Depressive episode (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Not related to vaccine
Elective caesarean section (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 2 (2) — Not related to vaccine
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Girls (1D Cervarix®) Systematic Collection Phase (N=620) | Women (3D Gardasil-4®) Systematic Collection Phase (N=620) | Girls (1D Cervarix®) Non-systematic Collection Phase (N=620) | Women (3D Gardasil-4®) Non-systematic Collection Phase (N=620)
Agranulocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Not related to vaccine
Anaemia, unspecified (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 4 (4) — Not related to vaccine. NOTE: Event was collected by both systematic and non-systematic methods.
Thrombocytopenia, unspecified (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Not related to vaccine
White blood cell disorder (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Not related to vaccine
Conduction disorder, unspecified (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Not related to vaccine
Pure hyperglyceridaemia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) — Not related to vaccine
Pure hypercholesterolaemia (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) — Not related to vaccine. NOTE: Event was collected by both systematic and non-systematic methods.
Hypopituitarism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Not related to vaccine
Thyroid disorder (Endocrine disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) — Not related to vaccine. NOTE: Event was collected by both systematic and non-systematic methods.
Myopia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Not related to vaccine
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Not related to vaccine
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Not related to vaccine
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Not related to vaccine
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Not related to vaccine
Irritable bowel (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Not related to vaccine
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Not related to vaccine
Tooth disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Not related to vaccine
Upper abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Not related to vaccine
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) — Not related to vaccine
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Probably related to vaccine
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Probably related to vaccine
Adverse drug reaction (General disorders) | 0 (0) | 3 (3) | 1 (1) | 2 (2) — Not related to vaccine. NOTE: Event was collected by both systematic and non-systematic methods.
Fever (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) — Not related to vaccine. NOTE: Event was collected by both systematic and non-systematic methods.
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Not related to vaccine
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Not related to vaccine
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Probably related to vaccine
Unspecified disorder of liver (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) — Not related to vaccine
Dengue (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) — Not related to vaccine. NOTE: Event was collected by both systematic and non-systematic methods.
Asthma, unspecified (Immune system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) — Not related to vaccine. NOTE: Event was collected by both systematic and non-systematic methods.
Allergy (Immune system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) — Not related to vaccine. NOTE: Event was collected by both systematic and non-systematic methods.
Allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Possibly related to vaccine
Allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Probably related to vaccine
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Not related to vaccine
Coronavirus disease 2019 (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 2 (2) — Not related to vaccine
Enterovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Not related to vaccine
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) — Not related to vaccine. NOTE: Event was collected by both systematic and non-systematic methods.
Gastrointestinal viral infection (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 0 (0) — Not related to vaccine
Genital herpes simplex (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) — Not related to vaccine
Impetigo (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Not related to vaccine
Influenza (Infections and infestations) | 5 (6) | 4 (4) | 9 (9) | 9 (9) — Not related to vaccine. NOTE: Event was collected by both systematic and non-systematic methods.
Papilloma viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Not related to vaccine
Sialoadenitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Not related to vaccine
Tinea corporis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Not related to vaccine
Unspecified otitis media (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Not related to vaccine
Urinary tract infection, site not specified (Infections and infestations) | 3 (3) | 12 (13) | 1 (1) | 4 (4) — Not related to vaccine. NOTE: Event was collected by both systematic and non-systematic methods.
Varicella (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — Not related to vaccine
Viral hepatitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Not related to vaccine
Viral infection (Infections and infestations) | 3 (3) | 8 (8) | 3 (3) | 5 (5) — Not related to vaccine. NOTE: Event was collected by both systematic and non-systematic methods.
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 3 (3) — Not related to vaccine
Acute nasopharyngitis (common cold) (Infections and infestations) | 8 (9) | 9 (9) | 2 (2) | 4 (4) — Not related to vaccine. NOTE: Event was collected by both systematic and non-systematic methods.
Acute upper respiratory tract infection (Infections and infestations) | 2 (2) | 6 (6) | 3 (3) | 0 (0) — Not related to vaccine. NOTE: Event was collected by both systematic and non-systematic methods.
Acute vaginitis (Infections and infestations) | 0 (0) | 3 (3) | 1 (1) | 0 (0) — Not related to vaccine. NOTE: Event was collected by both systematic and non-systematic methods.
Chronic ethmoidal sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Not related to vaccine
Laboratory confirmed COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 4 (4) | 7 (7) — Not related to vaccine. NOTE: Event was collected by both systematic and non-systematic methods.
Skin injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — Definitely related to vaccine
Breast injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Not related to vaccine
Burns second degree (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Not related to vaccine
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Not related to vaccine
Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Not related to vaccine
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Not related to vaccine
Musculoskeletal procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Not related to vaccine
Skin injury (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 0 (0) — Not related to vaccine
Trunk injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Not related to vaccine
Leg injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Not related to vaccine
Unspecified perineal laceration during delivery (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Not related to vaccine
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) — Not related to vaccine. NOTE: Event was collected by both systematic and non-systematic methods.
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) — Not related to vaccine. NOTE: Event was collected by both systematic and non-systematic methods.
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Definitely related to vaccine
Pain in limb (Musculoskeletal and connective tissue disorders) | 2 (2) | 10 (10) | 1 (1) | 0 (0) — Definitely related to vaccine. NOTE: Event was collected by both systematic and non-systematic methods.
Soft tissue disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Definitely related to vaccine
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Not related to vaccine
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — Not related to vaccine
Pain in joint (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Not related to vaccine
Pain in limb (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0) — Not related to vaccine
Soft tissue disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) — Not related to vaccine
Ankle sprain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Not related to vaccine
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Possibly related to vaccine
Pain in limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Possibly related to vaccine
Pain in limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) — Probably related to vaccine
Soft tissue disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Probably related to vaccine
Benign neoplasm of ovary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Not related to vaccine
Leiomyoma of uterus, unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Not related to vaccine
Venereal warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 2 (2) | 1 (1) — Not related to vaccine. NOTE: Event was collected by both systematic and non-systematic methods.
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — Definitely related to vaccine
Cerebral oedema (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Not related to vaccine
Pre-menstrual tension syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) — Not related to vaccine. NOTE: Event was collected by both systematic and non-systematic methods.
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Not related to vaccine
Headache (Nervous system disorders) | 1 (1) | 4 (4) | 0 (0) | 0 (0) — Not related to vaccine
Migraine, unspecified (Nervous system disorders) | 2 (2) | 2 (2) | 1 (1) | 1 (1) — Not related to vaccine. NOTE: Event was collected by both systematic and non-systematic methods.
Neuromyopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Not related to vaccine
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Not related to vaccine
Tension headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Not related to vaccine
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Possibly related to vaccine
Migraine, unspecified (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) — Possibly related to vaccine
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Probably related to vaccine
Headache (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) — Probably related to vaccine
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Not related to vaccine
Polyhydramnios (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Not related to vaccine
Threatened abortion (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 2 (2) — Not related to vaccine. NOTE: Event was collected by both systematic and non-systematic methods.
Opioid abuse (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Not related to vaccine
Somatization disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Not related to vaccine
Anxiety disorder (Psychiatric disorders) | 1 (1) | 5 (5) | 1 (1) | 1 (1) — Not related to vaccine. NOTE: Event was collected by both systematic and non-systematic methods.
Deliberate self-harm (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) — Not related to vaccine. NOTE: Event was collected by both systematic and non-systematic methods.
Delusional disorder, unspecified type (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Not related to vaccine
Depressive episode (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) — Not related to vaccine. NOTE: Event was collected by both systematic and non-systematic methods.
Emotional disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Not related to vaccine
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Not related to vaccine
Mixed anxiety and depressive disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Not related to vaccine
Anxiety disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Possibly related to vaccine
Panic disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Possibly related to vaccine
Unspecified urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Not related to vaccine
Menses irregular with excessive bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Not related to vaccine
Amenorrhoea (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) — Not related to vaccine
Cervical dysplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) — Not related to vaccine
Cervical uterine polyp (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Not related to vaccine
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 3 (3) | 1 (1) | 1 (1) — Not related to vaccine. NOTE: Event was collected by both systematic and non-systematic methods.
Dysplasia of cervix (uteri) (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) — Not related to vaccine. NOTE: Event was collected by both systematic and non-systematic methods.
Irregular menstruation (Reproductive system and breast disorders) | 0 (0) | 3 (3) | 1 (1) | 3 (3) — Not related to vaccine. NOTE: Event was collected by both systematic and non-systematic methods.
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) — Not related to vaccine. NOTE: Event was collected by both systematic and non-systematic methods.
Polycystic ovarian syndrome (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) — Not related to vaccine. NOTE: Event was collected by both systematic and non-systematic methods.
Polymenorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) — Not related to vaccine. NOTE: Event was collected by both systematic and non-systematic methods.
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — Not related to vaccine
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) — Not related to vaccine
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Not related to vaccine
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) — Not related to vaccine
Paraesthesia skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Definitely related to vaccine
Allergic contact dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) — Not related to vaccine
Chronic skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Not related to vaccine
Herpes simplex dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Not related to vaccine
Unspecified local infection of skin and subcutaneous tissue (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Not related to vaccine
Atopic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Not related to vaccine
Urticaria, unspecified (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Possibly related to vaccine
Abscesses of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Probably related to vaccine
Paraesthesia skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Probably related to vaccine
Skin hypoaesthesia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Probably related to vaccine
Sexual abuse (Social circumstances) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Not related to vaccine
Circulatory collapse (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) — Definitely related to vaccine
Per vaginal bleeding (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) — Not related to vaccine
Circulatory collapse (Vascular disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) — Not related to vaccine. NOTE: Event was collected by both systematic and non-systematic methods.
Essential hypertension (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) — Not related to vaccine. NOTE: Event was collected by both systematic and non-systematic methods.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2023-02-28): https://cdn.clinicaltrials.gov/large-docs/81/NCT03728881/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-28): https://cdn.clinicaltrials.gov/large-docs/81/NCT03728881/SAP_001.pdf